Version Date: April 8, 2013

NCI Protocol #: CITN06-ALT-803

**Local Protocol #:** CA-ALT-803-01-13

**TITLE:** A Phase 1/2 Study of the Clinical and Immunologic Effects of ALT-803, a Novel Recombinant IL-15 Complex in Patients with Advanced Melanoma

(Advanced Melanoma – ICD-10053571)

Sponsor: Altor BioScience

Hing C. Wong, Ph.D.

Altor Bioscience Corporation.

Miramar, Florida 33025

Telephone: 954-443-8600 Safety Data Fax: 954-443-8602

**Coordinating Center:** Cancer Immunotherapy Trials Network, Fred Hutchinson

Cancer Research Center

\*Principal Investigator: Kim Margolin, MD

University of Washington, Seattle Cancer Care Alliance

825 East Lake Ave E, G4810 Seattle WA 98109-1023 Telephone: 206-288-7341

Fax: 206-288-6681 kmargoli@seattlecca.org

Co-Investigators: Adil Daud, MD

University of California San Francisco

(415) 353-7392

adaud@medicine.ucsf.edu

Marc Ernstoff, MD

Dartmouth Hitchcock Medical Center

(603) 650-5534

marc.s.ernstoff@hitchcock.org

Thomas Waldmann, MD National Cancer Institute

(301) 496-6656

tawald@mail.nih.gov

NCI Protocol #:CITN06-ALT-803


# INVESTIGATOR SIGNATURE PAGE

| <b>Protocol Number:</b> | CA-ALT-803-01-13 |
|---|---|
| Protocol Title: | A Phase 1/2 Study of the Clinical and<br>Immunologic Effects of ALT-803, a Novel<br>Recombinant IL-15 Complex in Patients with<br>Advanced Melanoma |
| <b>Date of Protocol:</b><br>Version # 01 | April 8, 2013 |
| Sponsor Contact: | Alter BioScience |
| | Hing C. Wong, Ph.D. Altor Bioscience Corporation. Miramar, Florida 33025 Telephone: 954-443-8600 |
| | Safety Data Fax: 954-443-8602 |
| • • • | est that I have read, and that I understand and will abide by estrictions contained in the attached protocol. |
| Review Board (IRB), and I understa | s study without approval of the appropriate Institutional and that any changes in the protocol must be approved in in certain cases the FDA, before they can be implemented, nazards to subjects. |
| Principal Investigator's Signature | Date |
| Principal Investigator's Name (Print) | |


Statistician: Study Coordinator: N/A

Zoe Moodie, PhD Fred Hutchinson Cancer Research Center 1100 Fairview Ave N, Mail Stop M2-C200 Seattle, WA 98109 (206) 667-7077 Fax: (206) 667-4378

zoe@fhcrc.org

Responsible Research Nurse: N/A Responsible Data Manager: N/A

NCI-Supplied Agent(s): N/A

Other Agent(s): ALT-803: a "recombinant human superagonist interleukin-15 (IL-15) complex" (AKA, IL-15N72D:IL-15RαSu/IgG1 Fc complex) NSC#: TBD

| <b>Investigational Agent</b> | IND# | IND Sponsor |
|------------------------------|------|------------------------------|
| ALT-803 | TBD | Altor Bioscience Corporation |

**Protocol Type / Version # / Version Date:** Original/Version 1/April 8, 2013

NCI Protocol #:CITN06-ALT-803 Version Date: April 8, 2013

### **SCHEMA**

| | | Regimen D | escriptio | n | |
|---|---|---|---|---|---|
| Agent | Pre-Medications: Precautions | Dose | Route | Schedule | Cycle Length |
| ALT-803 | *1 dose of | 0.003 mg/kg | IV | D1, W1 | 42 days |
| | antipyretic medication within | or<br>0.006 mg/kg | | D1, W2 | (4 weeks on, 2 weeks off) With up to 4 cycles in the |
| | 30 min of ALT-803<br>administration | or<br>0.01 mg/kg<br>or | | D1, W3<br>D1, W4 | absence of unacceptable toxicity and disease |
| | *1 dose of<br>antipyretic<br>medication 4 h after | 0.02 mg/kg<br>or<br>0.03 mg/kg | | | progression |
| | ALT-803 administration | 0.03 mg/kg | | | |

<sup>\*</sup>Non-steroidal anti-inflammatory medication such as acetaminophen, ibuprofen, Naproxen or aspirin may be given per physician discretion. Not to exceed standard maximum thresholds:

Acetaminophen: not to exceed 3000 mg (3 g) in 24 hours

Ibuprofen: not to exceed 2400 mg in 24 hours Naproxen: not to exceed 1100 mg in 24 hours Aspirin: not to exceed 3800 mg in 24 hours

| | Dose Escalation Schedule |
|------------|----------------------------------------------------|
| Dose Level | Dose of ALT-803 |
| Level -1 | 0.001 mg/kg (only if the first level is too toxic) |
| Level 1 | 0.003 mg/kg |
| Level 2 | 0.006 mg/kg |
| Level 3 | 0.01 mg/kg |
| Level 4 | 0.02 mg/kg |
| Level 5 | 0.03 mg/kg |

NCI Protocol #:CITN06-ALT-803 Version Date: April 8, 2013

### 10. STUDY CALENDAR

Baseline evaluations are to be conducted within 1 to 30 days before start of protocol therapy, as indicated in the study calendar, except for pregnancy testing, which must be performed within 48 hours prior to initial ALT-803 administration. Scans and x-rays must be performed within 30 days before the start of therapy. In the event that the patient's condition is changing, laboratory evaluations should be repeated within 24 hours before initiating the next cycle of therapy. Please refer to the study calendar below for specific timing of required evaluations.

| | Pre-s | | | C | valo 1 ( | Waalsa) | | | F/U 14 days post last Cycle 2 (Weeks) injection | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | (scree | :mng)<br> | Cycle 1 (Weeks) W1 W2 W3 W4 W5 W6 | | | | | | W1 | W2 | injection | Visit | | | | |
| | Within 30 d | Within 14 d | D1 | D8 | D15 | D22 | D29 | D36 | D1 | D8 | W3<br>D15 | W4<br>D22 | W5<br>D29 | W6<br>D36 | | |
| ALT-803*(A) | | | X | X | X | X | | | X | X | X | X | | | | |
| Informed consent | X | | | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | | | | |
| Concomitant meds | X | | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Physical exam | | X | X | X | X | X | X | | X | X | X | X | X | | X | X |
| Vital signs | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Height | X | | | | | | | | | | | | | | | |
| Weight | X | X | X | | X | | X | X | X | X | | X | | X | X | X |
| Performance status | | X | X | | | | | | X | | | | | | X | X |
| CBC w/diff, plts | | X | X | X | X | X | X | | X | X | X | X | X | X | X | X |
| PT/PTT | | X | | | | | | | | | | | | | | |
| Serum chemistry <sup>a</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Antinuclear antibody (ANA) | X | | | | | | | | X | | | | | | | X |
| Electrocardiogram (ECG) <sup>b</sup> | | | X <sup>b</sup> X <sup>b</sup> | | | | | $X^{b}$ | X <sup>b</sup> X <sup>b</sup> | | | | | $X^{b}$ | | |
| ECHO (as indicated) | X | | | | | | | | 1 | | | | | | | |
| Adverse event evaluation | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Tumor measurements <sup>c</sup> | X | | ı | Tum | or meas | uremen | ts are re | peated | every 8 ± 1 | week a | nd 16 = | 2 weel | ks | | | X |

NCI Protocol #:CITN06-ALT-803


| CT, MRI, or PET of chest, | X | Documentation (radiologic) must be provided for patients removed from study for progressive disease. | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| abdomen, pelvis <sup>d</sup> CT or MRI Brain <sup>d</sup> [as indicated for symptoms only] | X | If negative at baseline, to be repeated only with symptoms | | | | | | | | | |
| Radiologic evaluation by RECIST 1.1 | X | Radiologic measurements should be performed every $8 \pm 1$ week and $16 \pm 2$ weeks | | | | | | | | | |
| B-HCG <sup>e</sup> | | X | | | | | | | | | |
| EBV serostatus | X | | | | | | | | | | |
| CMV serostatus | X | | | | | | | | | | |
| Thyroid studies: TSH, T4 | X | | | | | | | | | | X |
| PK | | X | | | | | X | | | | |
| WB Immunophenotyping <sup>g</sup> | | X | X | X | X | X | X | X | X | | |
| IFN-γ ELISPOT <sup>g</sup> | | X | | | | X | X | | X | | |
| NK-cell function <sup>g</sup> | | X | | | | X | X | | X | | |
| Plasma cytokines <sup>g</sup> | | X | | | | X | X | | X | | |
| Serum Ab to ALT-803 <sup>g</sup> | | X | | | | | X | | | X | |
| PBMC | | X | | | | X | X | | X | | X |
| Serum | | X | | | | X | X | | X | | |

Abbreviations: Ab, antibodies; CBC, complete blood count; CT, computed tomography; MRI, magnetic resonance imaging; NK, natural killer; PET, positron emission tomography; PK, pharmacokinetics; PPT, partial thromboplastin time; PT, prothrombin time

<sup>\*(</sup>A), Agent

<sup>&</sup>lt;sup>a</sup> Blood chemistries include: creatinine, glucose, total protein, blood urea nitrogen (BUN), total carbon dioxide (CO<sub>2</sub>), albumin, total bilirubin, phosphorus, alkaline phosphatase, aspartate transaminae (AST), and alanine transaminase (ALT)

<sup>&</sup>lt;sup>b</sup> ECGs are to be done before ALT-803 injections on Day 1 and 6 hours after the first ALT-803 injection (Day1) of all treatment cycles. In addition an ECG is to be done at the end of treatment, *i.e.*, end of cycle 1, or after subsequent cycles have been completed.

<sup>&</sup>lt;sup>c</sup> baseline tumor assessment scans should be done 1 to 30 days before beginning treatment.

<sup>&</sup>lt;sup>d</sup> CT, MRI, or PET is acceptable for imaging assessment purposes

<sup>&</sup>lt;sup>e</sup> Pregnancy test may be done up to 48 hours before ALT-803 administration

f See pharmacokinetic flow sheet for specific draw times

<sup>&</sup>lt;sup>g</sup> Blood for WB Immunophenotyping, IFN-γ ELISPOT, NK-cell function, plasma cytokines, and serum Ab to ALT-803 must be drawn **before** the patient receives ALT-803 injections on Days 1, 8, 15 and 22 of each treatment cycle.

Version Date: May 6, 2013

NCI Protocol #: CITN06-ALT-803

**Local Protocol #:** CA-ALT-803-01-13

**TITLE:** A Phase 1/2 Study of the Clinical and Immunologic Effects of ALT-803, a Novel Recombinant IL-15 Complex in Patients with Advanced Melanoma

(Advanced Melanoma – ICD-10053571)

Sponsor: Altor BioScience

Hing C. Wong, Ph.D.

Altor Bioscience Corporation.

Miramar, Florida 33025

Telephone: 954-443-8600 Safety Data Fax: 954-443-8602

**Coordinating Center:** Cancer Immunotherapy Trials Network, Fred Hutchinson

Cancer Research Center

\*Principal Investigator: Kim Margolin, MD

University of Washington, Seattle Cancer Care Alliance

825 East Lake Ave E, G4810 Seattle WA 98109-1023 Telephone: 206-288-7341

Fax: 206-288-6681 kmargoli@seattlecca.org

**Co-Investigators:** Adil Daud, MD

University of California San Francisco

(415) 353-7392

adaud@medicine.ucsf.edu

Marc Ernstoff, MD

Dartmouth Hitchcock Medical Center

(603) 650-5534

marc.s.ernstoff@hitchcock.org

Thomas Waldmann, MD National Cancer Institute

(301) 496-6656

tawald@mail.nih.gov

Version Date: May 6, 2013

# INVESTIGATOR SIGNATURE PAGE

| Protocol Number: | CA-ALT-803-01-13 |
|---|---|
| Protocol Title: | A Phase 1/2 Study of the Clinical and<br>Immunologic Effects of ALT-803, a Novel<br>Recombinant IL-15 Complex in Patients with<br>Advanced Melanoma |
| Date of Protocol:<br>Version # 01<br>Version # 02 | April 8, 2013<br>May 6, 2013 |
| Sponsor Contact: | Altor BioScience |
| | Hing C. Wong, Ph.D.<br>Altor Bioscience Corporation. |
| | Miramar, Florida 33025 |
| | Telephone: 954-443-8600<br>Safety Data Fax: 954-443-8602 |
| all the conditions, instructions, and read Additionally, I will not initiate this Review Board (IRB), and I understa | est that I have read, and that I understand and will abide by estrictions contained in the attached protocol. s study without approval of the appropriate Institutional and that any changes in the protocol must be approved in in certain cases the FDA, before they can be implemented, nazards to subjects. |
| Principal Investigator's Signature | Date |
| Principal Investigator's Name (Print) | |

Version Date: May 6, 2013

Statistician: Study Coordinator: N/A

Zoe Moodie, PhD Fred Hutchinson Cancer Research Center 1100 Fairview Ave N, Mail Stop M2-C200 Seattle, WA 98109 (206) 667-7077 Fax: (206) 667-4378

zoe@fhcrc.org

Responsible Research Nurse: N/A Responsible Data Manager: N/A

NCI-Supplied Agent(s): N/A

Other Agent(s): ALT-803: a "recombinant human superagonist interleukin-15 (IL-15) complex" (AKA, IL-15N72D:IL-15RαSu/IgG1 Fc complex) NSC#: TBD

| <b>Investigational Agent</b> | IND# | IND Sponsor |
|------------------------------|--------|------------------------------|
| ALT-803 | 118280 | Altor Bioscience Corporation |

**Protocol Type / Version # / Version Date:** Version 2/May 6, 2013

NCI Protocol #:CITN06-ALT-803 Version Date: May 6, 2013

### **SCHEMA**

| | | Regimen D | escriptio | n | |
|---|---|---|---|---|---|
| Agent | Pre-Medications: Precautions | Dose | Route | Schedule | Cycle Length |
| ALT-803 | *1 dose of | 0.003 mg/kg | IV | D1, W1 | 42 days |
| | antipyretic medication within | or<br>0.006 mg/kg | | D1, W2 | (4 weeks on, 2 weeks off) With up to 4 cycles in the |
| | 30 min of ALT-803<br>administration | or<br>0.01 mg/kg<br>or | | D1, W3<br>D1, W4 | absence of unacceptable toxicity and disease |
| | *1 dose of<br>antipyretic<br>medication 4 h after | 0.02 mg/kg<br>or<br>0.03 mg/kg | | | progression |
| | ALT-803 administration | 0.03 mg/kg | | | |

<sup>\*</sup>Non-steroidal anti-inflammatory medication including agents such as acetaminophen, ibuprofen, or Naproxen may be given per physician discretion. Not to exceed standard maximum thresholds, for example:

Acetaminophen: not to exceed 3000 mg (3 g) in 24 hours

Ibuprofen: not to exceed 2400 mg in 24 hours Naproxen: not to exceed 1100 mg in 24 hours

| | Dose Escalation Schedule |
|------------|----------------------------------------------------|
| Dose Level | Dose of ALT-803 |
| Level -1 | 0.001 mg/kg (only if the first level is too toxic) |
| Level 1 | 0.003 mg/kg |
| Level 2 | 0.006 mg/kg |
| Level 3 | 0.01 mg/kg |
| Level 4 | 0.02 mg/kg |
| Level 5 | 0.03 mg/kg |

NCI Protocol #:CITN06-ALT-803 Version Date: May 6, 2013

### 10. STUDY CALENDAR

Baseline evaluations are to be conducted within 1 to 30 days before start of protocol therapy, as indicated in the study calendar, except for pregnancy testing, which must be performed within 48 hours prior to initial ALT-803 administration. Scans and x-rays must be performed within 30 days before the start of therapy. In the event that the patient's condition is changing, laboratory evaluations should be repeated within 24 hours before initiating the next cycle of therapy. Please refer to the study calendar below for specific timing of required evaluations.

| | Pre-s | • | | | | | | | | | F/U 14<br>days post<br>last<br>injection | 6<br>Month<br>F/U<br>Visit | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | (scree | ening) | | | ycle 1 ( | | | | | Cy | injection | Visit | | | | |
| | Within 30 d | Within 14 d | W1<br>D1 | W2<br>D8 | W3<br>D15 | W4<br>D22 | W5<br>D29 | W6<br>D36 | W1<br>D1 | W2<br>D8 | W3<br>D15 | W4<br>D22 | W5<br>D29 | W6<br>D36 | | |
| ALT-803*(A) | | | X | X | X | X | | | X | X | X | X | | | | |
| Informed consent | X | | | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | | | | |
| Concomitant meds | X | | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Physical exam <sup>#</sup> | | X | X | X | X | X | X | | X | X | X | X | X | | X | X |
| Vital signs with oxygen saturation | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Height | X | | | | | | | | | | | | | | | |
| Weight | X | X | X | | X | | X | X | X | X | | X | | X | X | X |
| Performance status | | X | X | | | | | | X | | | | | | X | X |
| CBC w/diff, plts | | X | X | X | X | X | X | | X | X | X | X | X | X | X | X |
| PT/PTT | | X | | | | | | | | | | | | | | |
| Serum chemistry <sup>a</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Antinuclear antibody (ANA) | X | | | | | | | | X | | | | | | | X |
| Electrocardiogram (ECG) <sup>b</sup> | | | X <sup>b</sup> X <sup>b</sup> | | | | | $X^{b}$ | X <sup>b</sup> X <sup>b</sup> | | | | | $X^{b}$ | | |
| ECHO (as indicated) | X | | • | | | | | | | | | | | | | |
| Pulmonary function test (spirometry) | X | | | | | | | | | | | | | | | |

NCI Protocol #:CITN06-ALT-803


Version Date: May 6, 2013

| Adverse event evaluation | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Tumor measurements <sup>c</sup> | X | | I | Tum | or meas | uremen | ts are re | peated | every 8 ± 1 | week a | and 16 = | ± 2 weel | ks | | | X |
| CT, MRI, or PET of chest, abdomen, pelvis <sup>d</sup> | X | Doc | Documentation (radiologic) must be provided for patients removed from study for progressive disease. | | | | | | | | | | | | | |
| CT or MRI Brain <sup>d</sup> [as indicated for symptoms only] | X | | If negative at baseline, to be repeated only with symptoms | | | | | | | | | | | | | X |
| Radiologic evaluation by RECIST 1.1 | X | | Radiologic measurements should be performed every $8 \pm 1$ week and $16 \pm 2$ weeks | | | | | | | | | | | | | X |
| B-HCG <sup>e</sup> | | | X | | | | | | | | | | | | | |
| EBV serostatus | X | | | | | | | | | | | | | | | |
| CMV serostatus | X | | | | | | | | | | | | | | | |
| Thyroid studies: TSH, T4 | X | | | | | | | | | | | | | | | X |
| PK | | | X | | | | | | X | | | | | | | |
| WB Immunophenotyping <sup>g</sup> | | | X | X | X | X | X | | X | | X | | X | | | |
| IFN-γ ELISPOT <sup>g</sup> | | | X | | | | X | | X | | | | X | | | |
| NK-cell function <sup>g</sup> | | | X | | | | X | | X | | | | X | | | |
| Plasma cytokines <sup>g</sup> | | | X | | | | X | | X | | | | X | | | |
| Serum Ab to ALT-803 <sup>g</sup> | | | X | | | | | | X | | | | | | X | |
| PBMC | | | X | | | | X | | X | | | | X | | | X |
| Serum | | | X | | | | X | | X | | | | X | | | |

Abbreviations: Ab, antibodies; CBC, complete blood count; CT, computed tomography; MRI, magnetic resonance imaging; NK, natural killer; PET, positron emission tomography; PK, pharmacokinetics; PPT, partial thromboplastin time; PT, prothrombin time

<sup>\*(</sup>A), Agent

<sup>&</sup>lt;sup>#</sup> Physical exam must always include neurological assessment. In addition, all patients will have formal ophthalmologic testing prior to starting therapy and repeated if clinically indicated.

<sup>&</sup>lt;sup>a</sup> Blood chemistries include: creatinine, glucose, total protein, blood urea nitrogen (BUN), total carbon dioxide (CO<sub>2</sub>), albumin, total bilirubin, phosphorus, alkaline phosphatase, aspartate transaminase (AST), and alanine transaminase (ALT)

<sup>&</sup>lt;sup>b</sup> ECGs are to be done before ALT-803 injections on Day 1 and 4, 12 and 24 hours post-dose. ECGs are to be repeated before and at 4 hours (the end of the outpatient observation period) following each subsequent dose.

<sup>&</sup>lt;sup>c</sup> Baseline tumor assessment scans should be done 1 to 30 days before beginning treatment.

<sup>&</sup>lt;sup>d</sup> CT, MRI, or PET is acceptable for imaging assessment purposes

e Pregnancy test may be done up to 48 hours before ALT-803 administration

<sup>&</sup>lt;sup>f</sup> See pharmacokinetic flow sheet for specific draw times

<sup>&</sup>lt;sup>g</sup> Blood for WB Immunophenotyping, IFN-γ ELISPOT, NK-cell function, plasma cytokines, and serum Ab to ALT-803 must be drawn **before** the patient receives ALT-803 injections on Days 1, 8, 15 and 22 of each treatment cycle.

NCI Protocol #:CITN06-ALT-803

Version Date: July 26, 2013


NCI Protocol #: CITN06-ALT-803

**Local Protocol #:** CA-ALT-803-01-13

**TITLE:** A Phase 1/2 Study of the Clinical and Immunologic Effects of ALT-803, a Novel Recombinant IL-15 Complex in Patients with Advanced Melanoma

(Advanced Melanoma – ICD-10053571)

Sponsor: Altor BioScience

Hing C. Wong, Ph.D.

Altor Bioscience Corporation.

Miramar, Florida 33025

Telephone: 954-443-8600 Safety Data Fax: 954-443-8602

**Coordinating Center:** Cancer Immunotherapy Trials Network, Fred Hutchinson

Cancer Research Center

\*Principal Investigator: Kim Margolin, MD

University of Washington, Seattle Cancer Care Alliance

825 East Lake Ave E, G4810 Seattle WA 98109-1023 Telephone: 206-288-7341

Fax: 206-288-6681 kmargoli@seattlecca.org

**Co-Investigators:** Adil Daud, MD

University of California San Francisco

(415) 353-7392

adaud@medicine.ucsf.edu

Marc Ernstoff, MD

Dartmouth Hitchcock Medical Center

(603) 650-5534

marc.s.ernstoff@hitchcock.org

Thomas Waldmann, MD National Cancer Institute

(301) 496-6656

tawald@mail.nih.gov

# CONFIDENTIAL

Version Date: July 26, 2013

# INVESTIGATOR SIGNATURE PAGE

| <b>Protocol Number:</b> | CA-ALT-803-01-13 |
|---|---|
| Protocol Title: | A Phase 1/2 Study of the Clinical and<br>Immunologic Effects of ALT-803, a Novel<br>Recombinant IL-15 Complex in Patients with<br>Advanced Melanoma |
| Date of Protocol: | |
| Version # 01 | April 8, 2013 |
| Version # 02 | May 6, 2013 |
| Version # 03 | July 26, 2013 |
| Sponsor Contact: | Altor BioScience |
| | CORPORATION |
| | Hing C. Wong, Ph.D. |
| | Altor Bioscience Corporation. |
| | Miramar, Florida 33025 Telephone: 954-443-8600 |
| | Safety Data Fax: 954-443-8602 |
| | est that I have read, and that I understand and will abide by estrictions contained in the attached protocol. |
| Review Board (IRB), and I understa | s study without approval of the appropriate Institutional and that any changes in the protocol must be approved in in certain cases the FDA, before they can be implemented, hazards to subjects. |
| Principal Investigator's Signature | Date |
| Principal Investigator's Name (Print) | |

Version Date: July 26, 2013

Statistician: Study Coordinator: N/A

Zoe Moodie, PhD Fred Hutchinson Cancer Research Center 1100 Fairview Ave N, Mail Stop M2-C200 Seattle, WA 98109 (206) 667-7077 Fax: (206) 667-4378

zoe@fhcrc.org

Responsible Research Nurse: N/A Responsible Data Manager: N/A

NCI-Supplied Agent(s): N/A

Other Agent(s): ALT-803: a "recombinant human superagonist interleukin-15 (IL-15) complex" (AKA, IL-15N72D:IL-15RαSu/IgG1 Fc complex) NSC#: TBD

| <b>Investigational Agent</b> | IND# | IND Sponsor |
|------------------------------|--------|------------------------------|
| ALT-803 | 118280 | Altor Bioscience Corporation |

**Protocol Type / Version # / Version Date:** Version 3/July 26, 2013

NCI Protocol #:CITN06-ALT-803 Version Date: July 26, 2013

### **SCHEMA**

| | | Regimen D | escriptio | n | |
|---|---|---|---|---|---|
| Agent | Pre-Medications: Precautions | Dose | Route | Schedule | Cycle Length |
| ALT-803 | *1 dose of antipyretic medication within 30 min of ALT-803 administration *1 dose of antipyretic medication 4 h after ALT-803 administration | 0.001 mg/kg<br>or<br>0.003 mg/kg<br>or<br>0.006 mg/kg<br>or<br>0.01 mg/kg<br>or<br>0.02 mg/kg<br>or<br>0.03 mg/kg | IV | D1, W1<br>D1, W2<br>D1, W3<br>D1, W4 | 42 days (4 weeks on, 2 weeks off) With up to 4 cycles in the absence of unacceptable toxicity and disease progression |

<sup>\*</sup>Non-steroidal anti-inflammatory medication including agents such as acetaminophen, ibuprofen, or Naproxen may be given per physician discretion. Not to exceed standard maximum thresholds, for example:

Acetaminophen: not to exceed 3000 mg (3 g) in 24 hours

Ibuprofen: not to exceed 2400 mg in 24 hours Naproxen: not to exceed 1100 mg in 24 hours

| | <b>Dose Escalation Schedule</b> |
|------------|-----------------------------------------------------|
| Dose Level | Dose of ALT-803 |
| Level -1 | 0.0005 mg/kg (only if the first level is too toxic) |
| Level 1 | 0.001 mg/kg |
| Level 2 | 0.003 mg/kg |
| Level 3 | 0.006 mg/kg |
| Level 4 | 0.01 mg/kg |
| Level 5 | 0.02 mg/kg |
| Level 6 | 0.03 mg/kg |

NCI Protocol #:CITN06-ALT-803 Version Date: July 26, 2013

### 10. STUDY CALENDAR

Baseline evaluations are to be conducted within 1 to 30 days before start of protocol therapy, as indicated in the study calendar, except for pregnancy testing, which must be performed within 48 hours prior to initial ALT-803 administration. Scans and x-rays must be performed within 30 days before the start of therapy. In the event that the patient's condition is changing, laboratory evaluations should be repeated within 24 hours before initiating the next cycle of therapy. Please refer to the study calendar below for specific timing of required evaluations.

| | Pre-study | | | | ycle 1 ( | | | | | | | | | F/U 14<br>days post<br>last | 6<br>Month<br>F/U | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | (scree | ening) | **** | Cycle 2 (Weeks) | | | | | | injection | Visit | | | | | |
| | Within 30 d | Within 14 d | W1<br>D1 | W2<br>D8 | W3<br>D15 | W4<br>D22 | W5<br>D29 | W6<br>D36 | W1<br>D1 | W2<br>D8 | W3<br>D15 | W4<br>D22 | W5<br>D29 | W6<br>D36 | | |
| ALT-803*(A) | | | X | X | X | X | | | X | X | X | X | | | | |
| Informed consent | X | | | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | | | | |
| Concomitant meds | X | | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Physical exam <sup>#</sup> | | X | X | X | X | X | X | | X | X | X | X | X | | X | X |
| Vital signs with oxygen saturation | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Height | X | | | | | | | | | | | | | | | |
| Weight | X | X | X | | X | | X | X | X | X | | X | | X | X | X |
| Performance status | | X | X | | | | | | X | | | | | | X | X |
| CBC w/diff, plts | | X | X | X | X | X | X | | X | X | X | X | X | X | X | X |
| PT/PTT | | X | | | | | | | | | | | | | | |
| Serum chemistry <sup>a</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Antinuclear antibody (ANA) | X | | | | | | | | X | | | | | | | X |
| Electrocardiogram (ECG) <sup>b</sup> | | | X <sup>b</sup> X <sup>b</sup> | | | | | $X^{b}$ | X <sup>b</sup> X <sup>b</sup> | | | | | $X^{b}$ | | |
| ECHO (as indicated) | X | | • | | | | | | | | | | | | | |
| Pulmonary function test (spirometry) | X | | | | | | | | | | | | | | | |

NCI Protocol #:CITN06-ALT-803


Version Date: July 26, 2013

| Adverse event evaluation | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Tumor measurements <sup>c</sup> | X | | I | Tum | or meas | uremen | ts are re | peated | every 8 ± 1 | week a | and 16 = | 2 weel | ks | | | X |
| CT, MRI, or PET of chest, abdomen, pelvis <sup>d</sup> | X | Doc | Documentation (radiologic) must be provided for patients removed from study for progressive disease. | | | | | | | | | | | | se. | |
| CT or MRI Brain <sup>d</sup> [as indicated for symptoms only] | X | | If negative at baseline, to be repeated only with symptoms | | | | | | | | | | | X | | |
| Radiologic evaluation by RECIST 1.1 | X | | Rac | liologic | measur | ements | should | be perfo | ormed ever | y <u>8 ± 1</u> | week ai | nd 16 ± | 2 week | S | | X |
| B-HCG <sup>e</sup> | | | X | | | | | | | | | | | | | |
| EBV serostatus | X | | | | | | | | | | | | | | | |
| CMV serostatus | X | | | | | | | | | | | | | | | |
| Thyroid studies: TSH, T4 | X | | | | | | | | | | | | | | | X |
| PK | | | X | | | | | | X | | | | | | | |
| WB Immunophenotyping <sup>g</sup> | | | X | X | X | X | X | | X | | X | | X | | | |
| IFN-γ ELISPOT <sup>g</sup> | | | X | | | | X | | X | | | | X | | | |
| NK-cell function <sup>g</sup> | | | X | | | | X | | X | | | | X | | | |
| Plasma cytokines <sup>g</sup> | | | X | | | | X | | X | | | | X | | | |
| Serum Ab to ALT-803 <sup>g</sup> | | | X | | | | | | X | | | | | | X | |
| PBMC | | | X | | | | X | | X | | | | X | | | X |
| Serum | | | X | | | | X | | X | | | | X | | | |

Abbreviations: Ab, antibodies; CBC, complete blood count; CT, computed tomography; MRI, magnetic resonance imaging; NK, natural killer; PET, positron emission tomography; PK, pharmacokinetics; PPT, partial thromboplastin time; PT, prothrombin time

<sup>\*(</sup>A), Agen

<sup>&</sup>lt;sup>#</sup> Physical exam must always include neurological assessment. In addition, all patients will have formal ophthalmologic testing prior to starting therapy and repeated if clinically indicated.

<sup>&</sup>lt;sup>a</sup> Blood chemistries include: creatinine, glucose, total protein, blood urea nitrogen (BUN), total carbon dioxide (CO<sub>2</sub>), albumin, total bilirubin, phosphorus, alkaline phosphatase, aspartate transaminase (AST), and alanine transaminase (ALT)

<sup>&</sup>lt;sup>b</sup> ECGs are to be done before ALT-803 injections on Day 1 and 4, 12 and 24 hours post-dose. ECGs are to be repeated before and at 4 hours (the end of the outpatient observation period) following each subsequent dose.

<sup>&</sup>lt;sup>c</sup> Baseline tumor assessment scans should be done 1 to 30 days before beginning treatment.

<sup>&</sup>lt;sup>d</sup> CT, MRI, or PET is acceptable for imaging assessment purposes

e Pregnancy test may be done up to 48 hours before ALT-803 administration

<sup>&</sup>lt;sup>f</sup> See pharmacokinetic flow sheet for specific draw times

<sup>&</sup>lt;sup>g</sup> Blood for WB Immunophenotyping, IFN-γ ELISPOT, NK-cell function, plasma cytokines, and serum Ab to ALT-803 must be drawn **before** the patient receives ALT-803 injections on Days 1, 8, 15 and 22 of each treatment cycle.

Version Date: December 02, 2013

NCI Protocol #: CITN-06-ALT-803

**Local Protocol #:** CA-ALT-803-01-13

**TITLE:** A *Phase 1* Study of the Clinical and Immunologic Effects of ALT-803, a Novel Recombinant IL-15 Complex in Patients with Advanced Melanoma

(Advanced Melanoma – ICD-10053571)

Sponsor: Altor BioScience

Hing C. Wong, Ph.D.

Altor Bioscience Corporation. Miramar, Florida 33025

Telephone: 954-443-8600 Safety Data Fax: 954-443-8602

**Coordinating Center:** Cancer Immunotherapy Trials Network, Fred Hutchinson

Cancer Research Center

\*Principal Investigator: Kim Margolin, MD

University of Washington, Seattle Cancer Care Alliance

825 East Lake Ave E, G4810 Seattle WA 98109-1023 Telephone: 206-288-7341

Fax: 206-288-6681 kmargoli@seattlecca.org

**Co-Investigators:** Adil Daud, MD

University of California San Francisco

(415) 353-7392

adaud@medicine.ucsf.edu

Marc Ernstoff, MD

Dartmouth Hitchcock Medical Center

(603) 650-5534

marc.s.ernstoff@hitchcock.org

Thomas Waldmann, MD National Cancer Institute

(301) 496-6656

tawald@mail.nih.gov

The University of Washington and USCF will participate to the dose-escalation phase of the trial. Dartmouth and the NCI will be added in the expansion phase of the trial.

Version Date: December 02, 2013

# INVESTIGATOR SIGNATURE PAGE

| Protocol Number: | CA-ALT-803-01-13 |
|---|---|
| Protocol Title: | A <i>Phase 1</i> Study of the Clinical and Immunologic Effects of ALT-803, a Novel Recombinant IL-15 Complex in Patients with Advanced Melanoma |
| Date of Protocol: | |
| Version # 04 | December 02, 2013 |
| Sponsor Contact: | Altor BioScience |
| • | CORPORATION |
| | Hing C. Wong, Ph.D. |
| | Altor Bioscience Corporation. Miramar, Florida 33025 |
| | Telephone: 954-443-8600 |
| | Safety Data Fax: 954-443-8602 |
| all the conditions, instructions, and r<br>Additionally, I will not initiate th<br>Review Board (IRB), and I underst | test that I have read, and that I understand and will abide by estrictions contained in the attached protocol. is study without approval of the appropriate Institutional tand that any changes in the protocol must be approved in I, in certain cases the FDA, before they can be implemented, hazards to subjects. |
| Principal Investigator's Signature | |
| Principal Investigator's Name (Print | |

Version Date: December 02, 2013

Statistician: Study Coordinator: N/A

Zoe Moodie, PhD Fred Hutchinson Cancer Research Center 1100 Fairview Ave N, Mail Stop M2-C200 Seattle, WA 98109 (206) 667-7077 Fax: (206) 667-4378

Fax: (206) 667-4378 zoe@fhcrc.org

Responsible Research Nurse: N/A Responsible Data Manager: N/A

NCI-Supplied Agent(s): N/A

Other Agent(s): ALT-803: a "recombinant human superagonist interleukin-15 (IL-15) complex"

(AKA, IL-15N72D: IL-15RαSu/IgG1 Fc complex) NSC#: TBD

| <b>Investigational Agent</b> | IND# | IND Sponsor |
|------------------------------|--------|------------------------------|
| ALT-803 | 118280 | Altor Bioscience Corporation |

Protocol Type / Version # / Version Date: Amendment/Version 1.0/November 22, 2013

### CANCER TRIALS SUPPORT UNIT (CTSU) ADDRESS AND CONTACT INFORMATION

| To submit site registration documents: | For patient enrollments: | Submit study data |
|---|---|---|
| CTSU Regulatory Office 1818 Market Street, Suite 1100 Philadelphia, PA 19103 Phone – 1-866-651-CTSU Fax – 215-569-0206 Email: CTSURegulatory@ctsu.coccg.o rg (for submitting regulatory documents only) | Please refer to the patient enrollment section for instructions on using the Oncology Patient Enrollment Network (OPEN) at <a href="https://www.ctsu.org/OPEN_SYSTEM/">https://www.ctsu.org/OPEN_SYSTEM/</a> or <a href="https://OPEN.ctsu.org">https://OPEN.ctsu.org</a> . Contact the CTSU Help Desk with any OPEN-related questions at ctsucontact@westat.com. | Data collection for this study will be done via Medidata Rave (Axio Research). Please see the data submission section of the protocol for further instructions. |

The current version of the study protocol and all supporting documents must be downloaded from the protocol-specific Web page of the CTSU Member Web site located at <a href="https://www.ctsu.org">https://www.ctsu.org</a>.

For patient eligibility or treatment-related questions:

Contact the CITN Coordinating Center at <a href="mailto:citn@fhcrc.org">citn@fhcrc.org</a> or 206-667-6606

<u>For questions unrelated to patient eligibility, treatment, or clinical data submission</u> contact the CTSU Help Desk by phone or e-mail:

CTSU General Information Line – 1-888-823-5923, or <u>ctsucontact@westat.com</u>. All calls and correspondence will be triaged to the appropriate CTSU representative.

The CTSU Web site is located at <a href="https://www.ctsu.org">https://www.ctsu.org</a>

### **SCHEMA**

| | Regimen Description | | | | |
|---|---|---|---|---|---|
| Agent | Pre-Medications: Precautions | Dose | Route | Schedule | Cycle Length |
| ALT-803 | *1 dose of | <i>0.3 μg/kg</i> or | IV | D1, W1 | 42 days |
| | antipyretic medication within | 0.5 μg/kg or<br>1 μg/kg or | | D1, W2 | (4 weeks on, 2 weeks off) |
| | 30 min of ALT-803 | $3 \mu g/kg$ or | | D1, W3 | With up to 4 cycles in the absence of unacceptable |
| | administration | 6 μg/kg | | D1, W4 | toxicity and disease progression** |
| | *1 dose of | | | | progression |
| | antipyretic | | | | |
| | medication 4 h after | | | | |
| | ALT-803 | | | | |
| | administration | | | | |

<sup>\*</sup>Non-steroidal anti-inflammatory medication including agents such as acetaminophen, ibuprofen, or Naproxen may be given per physician discretion. Not to exceed standard maximum thresholds:

Acetaminophen: not to exceed 3000 mg (3 g) in 24 hours

Ibuprofen: not to exceed 2400 mg in 24 hours Naproxen: not to exceed 1100 mg in 24 hours

\*\* Additional cycles beyond the 4<sup>th</sup> cycle may be considered for patients continuing to benefit and tolerating therapy, upon discussion among the sponsor and Principal Investigator.

| | Dose Escalation Schedule |
|---|---|
| Dose Level | Dose of ALT-803 |
| Level -1 | $0.1 \mu g/kg$ (only if the first level is too toxic) |
| Level 1 | 0.3 μg/kg |
| Level 2 | $0.5 \mu g/kg$ |
| Level 3 | 1 μg/kg |
| Level 4 | 3 μg/kg |
| Level 5 | 6 μg/kg |

### 10. STUDY CALENDAR

Baseline evaluations are to be conducted within 1 to 30 days before start of protocol therapy, as indicated in the study calendar, except for pregnancy testing, which must be performed within 48 hours prior to initial ALT-803 administration. Scans and x-rays must be performed within 30 days before the start of therapy. In the event that the patient's condition is changing, laboratory evaluations should be repeated within 24 hours before initiating the next cycle of therapy. Please refer to the study calendar below for specific timing of required evaluations.

| | | | | | | | | | | | | | | | | F/U | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Pre-s<br>(scree | | | | Cycle 1 | (Weeks) | | | Cycle 2 (Weeks) | | | | | | 14 d<br>post<br>last inf. | 6<br>Mo | 1 year <sup>i</sup> |
| | Within | Within | W1 | W2 | W3 | W4 | W5 | W6 | W1 | W2 | W3 | W4 | W5 | W6 | | | • |
| ALT-803*(A) | 30 d | 14 d | D1±1<br>X | D8±1<br>X | D15±1<br>X | D22±1<br>X | D29±1 | D36±1 | D1± <i>1</i><br>X | D8±1<br>X | D15±1<br>X | D22±1<br>X | D29±1 | D36±1 | | | |
| Informed consent | X | | | | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | | | | | |
| Concomitant meds | X | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Physical exam <sup>h</sup> | | X | X | X | X | X | X | | X | X | X | X | X | | X | X | X |
| Vital signs with oxygen saturation | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Height | X | | | | | | | | | | | | | | | | |
| Weight | X | X | X | | X | | X | X | X | X | | X | | X | X | X | X |
| Performance status | | X | X | | | | | | X | | | | | | X | X | X |
| CBC w/diff, plts | | X | X | X | X | X | X | | X | X | X | X | X | X | X | X | X |
| PT/PTT | | X | | | | | | | | | | | | | | | |
| Serum chemistry <sup>a</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Antinuclear antibody (ANA) | X | | | | | | | | X | | | | | | | X | X |
| Electrocardiogram (ECG) <sup>b</sup> | | | X | X | X | X | | | X | X | X | X | | | X | X | X |
| ECHO (as indicated) | X | | | | | | | | | | | | | | | | |
| Adverse event evaluation | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Tumor measurements <sup>c</sup> CT, MRI, or PET of chest, | X<br>X | | Do | ocumenta | | | | | | | k and 12 ±<br>from stud | | ressive dis | sease. | 1 | X | |

NCI Protocol #:CITN-06-ALT-803


Version Date: December 02, 2013

| | | | | | | | | | | | | | F/U | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Pre-s<br>(scree | - | Cycle 1 (Weeks) | | | | | pos | | | | 14 d<br>post<br>last inf. | 6<br>Mo | 1 year <sup>i</sup> |
| abdomen, pelvis <sup>d</sup> | | | | | | | | | | | | | | |
| CT or MRI Brain <sup>d</sup> [as indicated for symptoms only] | X | | If negative at baseline, to be repeated only with symptoms | | | | | | | X | | | | |
| Radiologic evaluation by RECIST 1.1 | X | | Radiologic measurements should be performed every $6 \pm 1$ week and $12 \pm 2$ weeks | | | | | | X | | | | | |
| B-HCG <sup>e</sup> | | | X | | | | | | | | | | | |
| Thyroid studies: TSH, T4 | X | | | | | | | | | | | | X | X |
| $PK^f$ | | | X | | | | | | | | | | | |
| WB Immunophenotyping <sup>g</sup> | | | X | X | X | X | X | X | | X | X | | | |
| IFN-γ ELISPOT <sup>g</sup> | | | X | | | | X | X | | | X | | | |
| NK-cell function <sup>g</sup> | | | X | | | | X | X | | | X | | | |
| Plasma cytokines <sup>g</sup> | | | X | | | | X | X | | | X | | | |
| Serum Ab to ALT-803g | | | X | | | | | X | | | | X | | |
| Other laboratories <sup>j</sup> | | | X | | | | | | | | | | | |
| Serum | | | | | | | X | X | | | X | | | |

Abbreviations: Ab, antibodies; CBC, complete blood count; CT, computed tomography; MRI, magnetic resonance imaging; NK, natural killer; PET, positron emission tomography; PK, pharmacokinetics; *PTT*, partial thromboplastin time; PT, prothrombin time

<sup>\*(</sup>A), Agent

<sup>&</sup>lt;sup>a</sup> Blood chemistries include: creatinine, glucose, total protein, blood urea nitrogen (BUN), total carbon dioxide (CO<sub>2</sub>), albumin, total bilirubin, phosphorus, alkaline phosphatase, aspartate transaminase (AST), and alanine transaminase (ALT)

<sup>&</sup>lt;sup>b</sup> ECGs are to be done before ALT-803 infusions on Day 1 and 4, 12 and 24 hours after the first ALT-803 infusion (Cycle 1, Week 1, Day1). As clinically indicated, ECGs are to be obtained to evaluate for cardiac toxicity during subsequent doses and cycles of therapy and follow-up visits.

<sup>&</sup>lt;sup>c</sup> Baseline tumor assessment scans should be done 1 to 30 days before beginning treatment.

<sup>&</sup>lt;sup>d</sup> CT, MRI, or PET is acceptable for imaging assessment purposes

<sup>&</sup>lt;sup>e</sup> Pregnancy test may be done up to 48 hours before ALT-803 administration

f See pharmacokinetic flow sheet for specific draw times

<sup>&</sup>lt;sup>g</sup> Blood for WB Immunophenotyping, IFN-γ ELISPOT, NK-cell function, plasma cytokines, and serum Ab to ALT-803 must be drawn **before** the patient receives ALT-803 *infusions* on Days 1, 8, 15, and 22 of each treatment cycle.

h Physical exam must always include neurological assessment. In addition, all patients will have formal ophthalmologic testing prior to starting therapy and repeated if clinically indicated.

<sup>&</sup>lt;sup>1</sup>Additional cycles beyond the 4<sup>th</sup> cycle may be considered for patients continuing to benefit and tolerating therapy, upon discussion among the sponsor and Principal Investigator.

<sup>&</sup>lt;sup>j</sup>Other labs include: Lactate dehydrogenase, magnesium, phosphate, creatinine kinase and troponin I; must be drawn before and at 12 and 24 hours after the first ALT-803 dose.

NCI Protocol #: CITN-06-ALT-803

**Local Protocol #:** CA-ALT-803-01-13

**TITLE:** A Phase 1 Study of the Clinical and Immunologic Effects of ALT-803, a Novel Recombinant IL-15 Complex in Patients with Advanced Melanoma

(Advanced Melanoma – ICD-10053571)

Sponsor: Alter BioScience

Hing C. Wong, Ph.D.

Altor Bioscience Corporation.

Miramar, Florida 33025

Telephone: 954-443-8600 Safety Data Fax: 954-443-8602

**Coordinating Center:** Cancer Immunotherapy Trials Network, Fred Hutchinson

Cancer Research Center

\*Principal Investigator: Kim Margolin, MD

Stanford University, Division of Oncology

269 Campus Drive, CCSR 4115A

Stanford CA 94305-5151 kmargoli@stanford.edu

**Co-Investigators:** Adil Daud, MD

University of California San Francisco

(415) 353-7392

adaud@medicine.ucsf.edu

Lionel Lewis, MD

Dartmouth Hitchcock Medical Center

(603) 650-8685

lionel.lewis@dartmouth.edu

Sylvia Lee, MD

Seattle Cancer Care Alliance

(206) 667-2218 <u>smlee@fhcrc.org</u>

Shernan Holtan, MD University of Minnesota

(612) 301-1095 <u>sgholtan@umn.edu</u>

> Howard L. Kaufman, MD, FACS Rutgers University (732) 235-6807 Howard.kaufman@rutgers.edu

Thomas Waldmann, MD National Cancer Institute (301) 496-6656 tawald@mail.nih.gov

The SCCA, UCSF, Dartmouth, University of Minnesota, Rutgers University and Stanford University will participate to the dose-escalation phase of the trial. NCI will be added in the expansion phase of the trial.

## INVESTIGATOR SIGNATURE PAGE

| <b>Protocol Number:</b> | CA-ALT-803-01-13 |
|---|---|
| Protocol Title: | A Phase 1 Study of the Clinical and<br>Immunologic Effects of ALT-803, a Novel<br>Recombinant IL-15 Complex in Patients with<br>Advanced Melanoma |
| Date of Protocol: | |
| Version # 05 | October 08, 2014 |
| <b>Sponsor Contact:</b> | Alter BioScience |
| | Hing C. Wong, Ph.D. |
| | Altor Bioscience Corporation. |
| | Miramar, Florida 33025 |
| | Telephone: 954-443-8600 |
| | Safety Data Fax: 954-443-8602 |
| all the conditions, instructions, and Additionally, I will not initiate Review Board (IRB), and I under | attest that I have read, and that I understand and will abide by d restrictions contained in the attached protocol. this study without approval of the appropriate Institutional erstand that any changes in the protocol must be approved in and, in certain cases the FDA, before they can be implemented atte hazards to subjects. |
| Principal Investigator's Signature | Date |
| Principal Investigator's Name (Principal Investigator's Name ( | int) |

Statistician: Study Coordinator: N/A

Zoe Moodie, PhD Fred Hutchinson Cancer Research Center 1100 Fairview Ave N, Mail Stop M2-C200 Seattle, WA 98109 (206) 667-7077 Fax: (206) 667-4378 zoe@fhcrc.org

Responsible Research Nurse: N/A Responsible Data Manager: N/A

NCI-Supplied Agent(s): N/A

Other Agent(s): ALT-803: a "recombinant human superagonist interleukin-15 (IL-15) complex" (AKA, IL-15N72D: IL-15RαSu/IgG1 Fc complex) NSC#: TBD

| Investigational Agent | IND# | IND Sponsor |
|-----------------------|--------|------------------------------|
| ALT-803 | 118280 | Altor Bioscience Corporation |

Protocol Type / Version # / Version Date: Amendment / Version 3.0 / August 27, 2014

### CANCER TRIALS SUPPORT UNIT (CTSU) ADDRESS AND CONTACT INFORMATION

| To submit site registration | For patient enrollments: | Submit study data |
|---|---|---|
| documents: | | |
| CTSU Regulatory Office | Please refer to the patient enrollment | Data collection for this |
| 1818 Market Street, Suite 1100 | section for instructions on using the | study will be done via |
| Philadelphia, PA 19103 | Oncology Patient Enrollment Network | Medidata Rave (Axio |
| Phone – 1-866-651-CTSU | (OPEN) at | Research). |
| Fax – 215-569-0206 | https://www.ctsu.org/OPEN_SYSTEM/ | · |
| Email: | or <a href="https://OPEN.ctsu.org">https://OPEN.ctsu.org</a> . | Please see the data |
| CTSURegulatory@ctsu.coccg.o | | submission section of the |
| rg (for submitting regulatory | Contact the CTSU Help Desk with any | protocol for further |
| documents only) | OPEN-related questions at | instructions. |
| , | ctsucontact@westat.com. | |

The current version of the **study protocol and all supporting documents** must be downloaded from the protocol-specific Web page of the CTSU Member Web site located at <a href="https://www.ctsu.org">https://www.ctsu.org</a>.

### For patient eligibility or treatment-related questions:

Contact the CITN Coordinating Center at citn@fherc.org or 206-667-6606

For questions unrelated to patient eligibility, treatment, or clinical data submission contact the CTSU Help Desk by phone or e-mail:

CTSU General Information Line – 1-888-823-5923, or <a href="mailto:ctsucontact@westat.com">ctsucontact@westat.com</a>. All calls and correspondence will be triaged to the appropriate CTSU representative.

The CTSU Web site is located at <a href="https://www.ctsu.org">https://www.ctsu.org</a>

### **SCHEMA**

| | Regimen Description | | | | |
|---|---|---|---|---|---|
| Agent | Pre-Medications:<br>Precautions | Dose | Route | Schedule | Cycle Length |
| ALT-803 | *1 dose of | 0.3 μg/kg or | IV | D1, W1 | 42 days |
| | antipyretic medication within | 0.5 μg/kg or<br>1 μg/kg or | | D1, W2 | (4 weeks on, 2 weeks off) |
| | 30 min of ALT-803 | 3 μg/kg or | | D1, W3 | With up to 4 cycles in the |
| | administration 6 μg/kg | | | D1, W4 | absence of unacceptable toxicity and disease |
| | *1 dose of | | | | progression** |
| | antipyretic | | | | |
| | medication 4 h after | | | | |
| | ALT-803 | | | | |
| | administration | | | | |

<sup>\*</sup>Non-steroidal anti-inflammatory medication including agents such as acetaminophen, ibuprofen, or Naproxen may be given per physician discretion. Not to exceed standard maximum thresholds:

Acetaminophen: not to exceed 3000 mg (3 g) in 24 hours

Ibuprofen: not to exceed 2400 mg in 24 hours Naproxen: not to exceed 1100 mg in 24 hours

<sup>\*\*</sup> Additional cycles beyond the 4<sup>th</sup> cycle may be considered for patients continuing to benefit and tolerating therapy, upon discussion among the sponsor and Principal Investigator.

| | Dose Escalation Schedule |
|---|---|
| Dose Level | Dose of ALT-803 |
| Level -1 | 0.1 μg/kg (only if the first level is too toxic) |
| Level 1 | 0.3 μg/kg |
| Level 2 | 0.5 μg/kg |
| Level 3 | 1 μg/kg |
| Level 4 | 3 μg/kg |
| Level 5 | 6 μg/kg |

### 10. STUDY CALENDAR

Baseline evaluations are to be conducted within 1 to 30 days before start of protocol therapy, as indicated in the study calendar, except for pregnancy testing, which must be performed within 48 hours prior to initial ALT-803 administration. Scans and x-rays must be performed within 30 days before the start of therapy. In the event that the patient's condition is changing, laboratory evaluations should be repeated within 24 hours before initiating the next cycle of therapy. Please refer to the study calendar below for specific timing of required evaluations.

| | | 1. | | | | | | | | | | | | | | F/U | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Pre-s<br>(scree | | | | Cycle 1 | (Weeks) | | | Cycle 2 (Weeks) | | | | | | 14 d<br>post<br>last inf. | 6<br>Mo | 1 year <sup>i</sup> |
| | Within 30 d | Within<br>14 d | W1<br>D1±1 | W2<br>D8±1 | W3<br>D15±1 | W4<br>D22±1 | W5<br>D29±1 | W6<br>D36±1 | W1<br>D1±1 | W2<br>D8±1 | W3<br>D15±1 | W4<br>D22±1 | W5<br>D29±1 | W6<br>D36±1 | last IIII. | 1410 | 1 year |
| ALT-803*(A) | | | X | X | X | X | | | X | X | X | X | | | | | |
| Informed consent | X | | | | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | | | | | |
| Concomitant meds | X | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Physical exam <sup>h</sup> | | X | X | X | X | X | X | | X | X | X | X | X | | X | X | X |
| Vital signs with oxygen saturation | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Height | X | | | | | | | | | | | | | | | | |
| Weight | X | X | X | | X | | X | X | X | X | | X | | X | X | X | X |
| Performance status | | X | X | | | | | | X | | | | | | X | X | X |
| CBC w/diff, plts | | X | $X^k$ | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| PT/PTT | | X | | | | | | | | | | | | | | | |
| Serum chemistry <sup>a</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Antinuclear antibody (ANA) | X | | | | | | | | X | | | | | | | X | X |
| Electrocardiogram (ECG) <sup>b</sup> | | | X | X | X | X | | | X | X | X | X | | | X | X | X |
| ECHO (as indicated) | X | | | | | | | | | | | | | | | | |
| Adverse event evaluation | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Tumor measurements <sup>c</sup> CT, MRI, or PET of chest, abdomen, pelvis <sup>d</sup> | X<br>X | | Tumor measurements are repeated every $6 \pm 1$ week and $12 \pm 2$ weeks Documentation (radiologic) must be provided for patients removed from study for progressive disease. | | | | | | | | X | | | | | | |
| CT or MRI Brain <sup>d</sup> [as indicated for sympt only] | X | | If negative at baseline, to be repeated only with symptoms | | | | | | | | | X | | | | | |

| | | | | | | | | | | | | | | | | F/U | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Pre-s<br>(scree | · | Cycle 1 (Weeks) | | | | | | | Cycle 2 (Weeks) | | | | | | 6<br>Mo | 1 year <sup>i</sup> |
| | Within | Within | W1 | W2 | W3 | W4 | W5 | W6 | W1 | W2 | W3 | W4 | W5 | W6 | last inf. | 1710 | 1 year |
| | 30 d | 14 d | D1±1 | D8±1 | D15±1 | D22±1 | D29±1 | D36±1 | D1±1 | | D15±1 | D22±1 | D29±1 | D36±1 | | | |
| Radiologic evaluation by RECIST 1.1 | X | | Radiologic measurements should be performed every $6 \pm 1$ week and $12 \pm 2$ weeks | | | | | | | | | | X | | | | |
| B-HCG <sup>e</sup> | | | X | | | | | | | | | | | | | | |
| Thyroid studies: TSH, T4 | X | | | | | | | | | | | | | | | X | X |
| PK <sup>f</sup> | | | X | | | | | | | | | | | | | | |
| WB Immunophenotyping <sup>g</sup> | | | X | X | X | X | X | | X | | X | | X | | | | |
| IFN-γ ELISPOT <sup>g</sup> | | | X | | | | X | | X | | | | X | | | | |
| NK-cell function <sup>g</sup> | | | X | | | | X | | X | | | | X | | | | |
| Plasma cytokines <sup>g</sup> | | | X | | | | X | | X | | | | X | | | | |
| Kyn/Trp ratio <sup>g</sup> | | | X | | | | X | | X | | | | X | | | | |
| Serum Ab to ALT-803 <sup>g</sup> | | | X | | | | | | X | | | | | | X | | |
| Other laboratories <sup>j</sup> | | | X | | | | | | | | | | | | | | |
| Serum | | | | | | | X | | X | | | | X | | | | |

Abbreviations: Ab, antibodies; CBC, complete blood count; CT, computed tomography; MRI, magnetic resonance imaging; NK, natural killer; PET, positron emission tomography; PK, pharmacokinetics; PTT, partial thromboplastin time; PT, prothrombin time

<sup>\*(</sup>A): Agent

<sup>&</sup>lt;sup>a</sup> Blood chemistries include: creatinine, glucose, total protein, blood urea nitrogen (BUN), total carbon dioxide (CO<sub>2</sub>), albumin, total bilirubin, phosphorus, alkaline phosphatase, aspartate transaminase (AST), and alanine transaminase (ALT)

<sup>&</sup>lt;sup>b</sup> ECGs are to be done before ALT-803 infusions on Day 1 and 4, 12 and 24 hours after the first ALT-803 infusion (Cycle 1, Week 1, Day1). As clinically indicated, ECGs are to be obtained to evaluate for cardiac toxicity during subsequent doses and cycles of therapy and follow-up visits.

<sup>&</sup>lt;sup>c</sup> Baseline tumor assessment scans should be done 1 to 30 days before beginning treatment.

<sup>&</sup>lt;sup>d</sup> CT, MRI, or PET is acceptable for imaging assessment purposes

<sup>&</sup>lt;sup>e</sup> Pregnancy test may be done up to 48 hours before ALT-803 administration

See pharmacokinetic flow sheet for specific draw times

<sup>&</sup>lt;sup>g</sup> Blood for WB Immunophenotyping, IFN-γ ELISPOT, NK-cell function, plasma cytokines, *Kyn/Trp ratio* and serum Ab to ALT-803 must be drawn **before** the patient receives ALT-803 infusions on Days 1, 8, 15, and 22 of each treatment cycle.

h Physical exam must always include neurological assessment. In addition, a funduscopic exam, conducted by the investigator with a hand-held ophthalmoscope, must be done prior to starting therapy (Cycle 1, Day 1, Week 1) and repeated if clinically indicated (See Section 6.0 for additional details).

<sup>&</sup>lt;sup>1</sup>Additional cycles beyond the 4<sup>th</sup> cycle may be considered for patients continuing to benefit and tolerating therapy, upon discussion among the sponsor and Principal Investigator. <sup>j</sup>Other labs include: Lactate dehydrogenase, magnesium, phosphate, CK and troponin *I or T*; must be drawn **before** and at 12 and 24 hours after the first ALT-803 dose.

<sup>\*</sup>CBC w/diff, plts (Cycle 1, Week 1, Day 1); must be drawn before and at 12 and 24 hours after the first ALT-803 dose.

NCI Protocol #: CITN-06-ALT-803

**Local Protocol #:** CA-ALT-803-01-13

TITLE: A Phase 1 Study of the Clinical and Immunologic Effects of ALT-803, a Novel Recombinant IL-15 Complex in Patients with Advanced *Solid Tumors: Melanoma, Renal Cell, Non-Small Cell Lung and Squamous Cell Head and Neck Cancer* 

Sponsor: Alter BioScience

Hing C. Wong, Ph.D.

Altor Bioscience Corporation. Miramar, Florida 33025

Telephone: 954-443-8600 Safety Data Fax: 954-443-8602

**Coordinating Center:** Cancer Immunotherapy Trials Network, Fred Hutchinson

Cancer Research Center

\*Principal Investigator: Kim Margolin, MD

Stanford University, Division of Oncology

269 Campus Drive, CCSR 4115A

Stanford CA 94305-5151

(650) 725-5421

kmargoli@stanford.edu

Co-Investigators: Lionel Lewis, MD

Dartmouth Hitchcock Medical Center

(603) 650-8685

lionel.lewis@dartmouth.edu

Sylvia Lee, MD

Seattle Cancer Care Alliance

(206) 667-2218 smlee@fhcrc.org

Shernan Holtan, MD University of Minnesota

(612) 301-1095 <u>sgholtan@umn.edu</u>

> Howard L. Kaufman, MD, FACS Rutgers University (732) 235-6807 Howard.kaufman@rutgers.edu

Marc Ernstoff, MD Cleveland Clinic Foundation (216) 444-0888 ernstom@ccf.org

Thomas Waldmann, MD National Cancer Institute (301) 496-6656 tawald@mail.nih.gov

The SCCA, *Cleveland Clinic Foundation*, UCSF, Dartmouth, University of Minnesota, Rutgers University and Stanford University will participate to the dose-escalation phase of the trial. NCI will be added in the expansion phase of the trial.

# INVESTIGATOR SIGNATURE PAGE

| <b>Protocol Number:</b> | CA-ALT-803-01-13 |
|---|---|
| Protocol Title: | A Phase 1 Study of the Clinical and Immunologic Effects of ALT-803, a Novel Recombinant IL-15 Complex in Patients with Advanced <i>Solid Tumors:</i> Melanoma, <i>Renal Cell, Non-Small Cell Lung and Squamous Cell Head and Neck Cancer</i> |
| Date of Protocol: | |
| Version # 05 | October 08, 2014 |
| Version # 06 | November 20, 2014 |
| Sponsor Contact: | Altor BioScience |
| | Hing C. Wong, Ph.D. |
| | Altor Bioscience Corporation. |
| | Miramar, Florida 33025 |
| | Telephone: 954-443-8600 |
| | Safety Data Fax: 954-443-8602 |
| all the conditions, instructions, and Additionally, I will not initiate Review Board (IRB), and I und | attest that I have read, and that I understand and will abide by ad restrictions contained in the attached protocol. this study without approval of the appropriate Institutional erstand that any changes in the protocol must be approved in and, in certain cases the FDA, before they can be implemented, |
| except where necessary to elimin | |
| Principal Investigator's Signature | Date |
| Principal Investigator's Name (Pr | rint) |
Statistician: Study Coordinator: N/A

Zoe Moodie, PhD Fred Hutchinson Cancer Research Center 1100 Fairview Ave N, Mail Stop M2-C200 Seattle, WA 98109 (206) 667-7077 Fax: (206) 667-4378

zoe@fhcrc.org

Responsible Research Nurse: N/A Responsible Data Manager: N/A

NCI-Supplied Agent(s): N/A

Other Agent(s): ALT-803: a "recombinant human superagonist interleukin-15 (IL-15) complex" (AKA, IL-15N72D: IL-15RαSu/IgG1 Fc complex) NSC#: TBD

| <b>Investigational Agent</b> | IND# | IND Sponsor |
|------------------------------|--------|------------------------------|
| ALT-803 | 118280 | Altor Bioscience Corporation |

Protocol Type / Version # / Version Date: Amendment / Version 4.0 / October 30, 2014

### CANCER TRIALS SUPPORT UNIT (CTSU) ADDRESS AND CONTACT INFORMATION

| To submit site registration | For patient enrollments: | Submit study data |
|---|---|---|
| documents: | | |
| CTSU Regulatory Office | Please refer to the patient enrollment | Data collection for this |
| 1818 Market Street, Suite 1100 | section for instructions on using the | study will be done via |
| Philadelphia, PA 19103 | Oncology Patient Enrollment Network | Medidata Rave (Axio |
| Phone – 1-866-651-CTSU | (OPEN) at | Research). |
| Fax – 215-569-0206 | https://www.ctsu.org/OPEN_SYSTEM/ | |
| Email: | or <a href="https://OPEN.ctsu.org">https://OPEN.ctsu.org</a> . | Please see the data |
| CTSURegulatory@ctsu.coccg.o | | submission section of the |
| rg (for submitting regulatory | Contact the CTSU Help Desk with any | protocol for further |
| documents only) | OPEN-related questions at | instructions. |
| | ctsucontact@westat.com. | |

The current version of the **study protocol and all supporting documents** must be downloaded from the protocol-specific Web page of the CTSU Member Web site located at <a href="https://www.ctsu.org">https://www.ctsu.org</a>.

# For patient eligibility or treatment-related questions:

Contact the CITN Coordinating Center at citn@fherc.org or 206-667-6606

For questions unrelated to patient eligibility, treatment, or clinical data submission contact the CTSU Help Desk by phone or e-mail:

CTSU General Information Line – 1-888-823-5923, or <u>ctsucontact@westat.com</u>. All calls and correspondence will be triaged to the appropriate CTSU representative.

The CTSU Web site is located at <a href="https://www.ctsu.org">https://www.ctsu.org</a>

### **SCHEMA**

| | Regimen Description | | | | |
|---|---|---|---|---|---|
| Agent | Pre-Medications: Precautions | Dose | Route | Schedule | Cycle Length |
| ALT-803 | *1 dose of | 0.3 μg/kg or | IV | D1, W1 | 42 days |
| | antipyretic<br>medication within<br>30 min of ALT-803 | 0.5 μg/kg or<br>1 μg/kg or<br>3 μg/kg or | | D1, W2<br>D1, W3 | (4 weeks on, 2 weeks off) With up to 4 cycles in the absence of unacceptable |
| | administration *1 dose of | 6 μg/kg | | D1, W4 | toxicity and disease progression** |
| | antipyretic<br>medication 4 h after<br>ALT-803 | | | | |
| | administration | | | | |

<sup>\*</sup>Non-steroidal anti-inflammatory medication including agents such as acetaminophen, ibuprofen, or Naproxen may be given per physician discretion. Not to exceed standard maximum thresholds:

Acetaminophen: not to exceed 3000 mg (3 g) in 24 hours

Ibuprofen: not to exceed 2400 mg in 24 hours Naproxen: not to exceed 1100 mg in 24 hours

<sup>\*\*</sup> Additional cycles beyond the 4<sup>th</sup> cycle may be considered for patients continuing to benefit and tolerating therapy, upon discussion among the sponsor and Principal Investigator.

| | Dose Escalation Schedule |
|------------|--------------------------------------------------|
| Dose Level | Dose of ALT-803 |
| Level -1 | 0.1 μg/kg (only if the first level is too toxic) |
| Level 1 | 0.3 μg/kg |
| Level 2 | 0.5 μg/kg |
| Level 3 | 1 μg/kg |
| Level 4 | 3 μg/kg |
| Level 5 | 6 μg/kg |

### 10. STUDY CALENDAR

Baseline evaluations are to be conducted within 1 to 30 days before start of protocol therapy, as indicated in the study calendar, except for pregnancy testing, which must be performed within 48 hours prior to initial ALT-803 administration. Scans and x-rays must be performed within 30 days before the start of therapy. In the event that the patient's condition is changing, laboratory evaluations should be repeated within 24 hours before initiating the next cycle of therapy. Please refer to the study calendar below for specific timing of required evaluations.

| | | 1. | | | | | | | 1 | | | | | | | F/U | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | } | | | | | | | | | | | | 14 d | F/U | |
| | Pre-s<br>(scree | | | | Cycle 1 | (Weeks) | | | | | Cycle 2 | 2 (Weeks) | ) | | post<br>last inf. | 6<br>Mo | 1 year <sup>i</sup> |
| | Within 30 d | Within<br>14 d | W1<br>D1±1 | W2<br>D8±1 | W3<br>D15±1 | W4<br>D22±1 | W5<br>D29±1 | W6<br>D36±1 | W1<br>D1±1 | W2<br>D8±1 | W3<br>D15±1 | W4<br>D22±1 | W5<br>D29±1 | W6<br>D36±1 | | | |
| ALT-803*(A) | | | X | X | X | X | | | X | X | X | X | | | | | |
| Informed consent | X | | | | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | | | | | |
| Concomitant meds | X | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Physical exam <sup>h</sup> | | X | X | X | X | X | X | | X | X | X | X | X | | X | X | X |
| Vital signs with oxygen saturation | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Height | X | | | | | | | | | | | | | | | | |
| Weight | X | X | X | | X | | X | X | X | X | | X | | X | X | X | X |
| Performance status | | X | X | | | | | | X | | | | | | X | X | X |
| CBC w/diff, plts | | X | $X^k$ | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| PT/PTT | | X | | | | | | | | | | | | | | | |
| Serum chemistry <sup>a</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Antinuclear antibody (ANA) | X | | | | | | | | X | | | | | | | X | X |
| Electrocardiogram (ECG) <sup>b</sup> | | | X | X | X | X | | | X | X | X | X | | | X | X | X |
| ECHO (as indicated) | X | | | | | | | | | | | | | | | | |
| Adverse event evaluation | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Tumor measurements <sup>c</sup> | X | | Tumor measurements are repeated every $6 \pm 1$ week and $12 \pm 2$ weeks | | | | | | | | | | X | | | | |
| CT, MRI, or PET of chest, abdomen, pelvis <sup>d</sup> | X | | Do | ocumenta | ition (radi | - ' | | | | | from stud | | ressive dis | sease. | | | |
| CT or MRI Brain <sup>d</sup> [as indicated for sympt only] | X | | | | | If negati | ve at base | eline, to be | e repeate | d only w | ith sympto | oms | | | | X | |

| | | | | | | | | | | | | | | | | F/U | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Pre-s<br>(scree | | | | | | | | Cycle 2 (Weeks) | | | | | | 14 d<br>post<br>last inf. | 6<br>Mo | 1 year <sup>i</sup> |
| | Within | Within | W1 | W2 | W3 | W4 | W5 | W6 | W1 | W2 | W3 | W4 | W5 | W6 | last IIII. | 1710 | 1 year |
| | 30 d | 14 d | D1±1 | D8±1 | D15±1 | D22±1 | D29±1 | D36±1 | D1±1 | D8±1 | D15±1 | D22±1 | D29±1 | D36±1 | | | |
| Radiologic evaluation by RECIST 1.1 | X | | | R | adiologic | measuren | nents sho | uld be per | formed e | every 6 ± | 1 week ar | $12 \pm 2$ | weeks | | | X | |
| B-HCG <sup>e</sup> | | | X | | | | | | | | | | | | | | |
| Thyroid studies: TSH, T4 | X | | | | | | | | | | | | | | | X | X |
| PK <sup>f</sup> | | | X | | | | | | | | | | | | | | |
| WB Immunophenotyping <sup>g</sup> | | | X | X | X | X | X | | X | | X | | X | | | | |
| IFN-γ ELISPOT <sup>g</sup> | | | X | | | | X | | X | | | | X | | | | |
| NK-cell function <sup>g</sup> | | | X | | | | X | | X | | | | X | | | | |
| Plasma cytokines <sup>g</sup> | | | X | | | | X | | X | | | | X | | | | |
| Kyn/Trp ratio <sup>g</sup> | | | X | | | | X | | X | | | | X | | | | |
| Serum Ab to ALT-803 <sup>g</sup> | | | X | | | | | | X | | | | | | X | | |
| Other laboratories <sup>j</sup> | | | X | | | | | | | | | | | | | | |
| Serum | | | | | | | X | | X | | | | X | | | | |

Abbreviations: Ab, antibodies; CBC, complete blood count; CT, computed tomography; MRI, magnetic resonance imaging; NK, natural killer; PET, positron emission tomography; PK, pharmacokinetics; PTT, partial thromboplastin time; PT, prothrombin time

<sup>\*(</sup>A): Agent

<sup>&</sup>lt;sup>a</sup> Blood chemistries include: creatinine, glucose, total protein, blood urea nitrogen (BUN), total carbon dioxide (CO<sub>2</sub>), albumin, total bilirubin, phosphorus, alkaline phosphatase, aspartate transaminase (AST), and alanine transaminase (ALT)

<sup>&</sup>lt;sup>b</sup> ECGs are to be done before ALT-803 infusions on Day 1 and 4, 12 and 24 hours after the first ALT-803 infusion (Cycle 1, Week 1, Day1). As clinically indicated, ECGs are to be obtained to evaluate for cardiac toxicity during subsequent doses and cycles of therapy and follow-up visits.

<sup>&</sup>lt;sup>c</sup> Baseline tumor assessment scans should be done 1 to 30 days before beginning treatment.

<sup>&</sup>lt;sup>d</sup> CT, MRI, or PET is acceptable for imaging assessment purposes

<sup>&</sup>lt;sup>e</sup> Pregnancy test may be done up to 48 hours before ALT-803 administration

f See pharmacokinetic flow sheet for specific draw times

<sup>&</sup>lt;sup>g</sup> Blood for WB Immunophenotyping, IFN-γ ELISPOT, NK-cell function, plasma cytokines, Kyn/Trp ratio and serum Ab to ALT-803 must be drawn **before** the patient receives ALT-803 infusions on Days 1, 8, 15, and 22 of each treatment cycle.

h Physical exam must always include neurological assessment. In addition, a funduscopic exam, conducted by the investigator with a hand-held ophthalmoscope, must be done prior to starting therapy (Cycle 1, Day 1, Week 1) and repeated if clinically indicated (See Section 6.0 for additional details).

<sup>&</sup>lt;sup>1</sup>Additional cycles beyond the 4<sup>th</sup> cycle may be considered for patients continuing to benefit and tolerating therapy, upon discussion among the sponsor and Principal Investigator. <sup>j</sup>Other labs include: Lactate dehydrogenase, magnesium, phosphate, CK and troponin I or T; must be drawn **before** and at 12 and 24 hours after the first ALT-803 dose. <sup>k</sup>CBC w/diff, plts (Cycle 1, Week 1, Day 1); must be drawn **before** and at **12** and **24** hours after the first ALT-803 dose.

NCI Protocol #: CITN-06-ALT-803

**Local Protocol #:** CA-ALT-803-01-13

**TITLE:** A Phase 1 Study of the Clinical and Immunologic Effects of ALT-803, a Novel Recombinant IL-15 Complex in Patients with Advanced Solid Tumors: Melanoma, Renal Cell, Non-Small Cell Lung and Squamous Cell Head and Neck Cancer

Sponsor: Alter BioScience

Hing C. Wong, Ph.D.

Altor Bioscience Corporation.

Miramar, Florida 33025

Telephone: 954-443-8600 Safety Data Fax: 954-443-8602

**Coordinating Center:** Cancer Immunotherapy Trials Network, Fred Hutchinson

Cancer Research Center

\*Principal Investigator: Kim Margolin, MD

Stanford University, Division of Oncology

269 Campus Drive, CCSR 4115A

Stanford CA 94305-5151

(650) 725-5421

kmargoli@stanford.edu

Co-Investigators: Lionel Lewis, MD

Dartmouth Hitchcock Medical Center

(603) 650-8685

lionel.lewis@dartmouth.edu

Sylvia Lee, MD

Seattle Cancer Care Alliance

(206) 667-2218 smlee@fhcrc.org

Shernan Holtan, MD University of Minnesota

(612) 301-1095 <u>sgholtan@umn.edu</u>

> Howard L. Kaufman, MD, FACS Rutgers University (732) 235-6807 Howard.kaufman@rutgers.edu

Marc Ernstoff, MD Cleveland Clinic Foundation (216) 444-0888 ernstom@ccf.org

Thomas Waldmann, MD National Cancer Institute (301) 496-6656 tawald@mail.nih.gov

The SCCA, Cleveland Clinic Foundation, UCSF, Dartmouth, University of Minnesota, Rutgers University and Stanford University will participate to the dose-escalation phase of the trial. NCI will be added in the expansion phase of the trial.

# INVESTIGATOR SIGNATURE PAGE

| <b>Protocol Number:</b> | CA-ALT-803-01-13 |
|---|---|
| Protocol Title: | A Phase 1 Study of the Clinical and<br>Immunologic Effects of ALT-803, a Novel<br>Recombinant IL-15 Complex in Patients with<br>Advanced Solid Tumors: Melanoma, Renal Cell,<br>Non-Small Cell Lung and Squamous Cell Head<br>and Neck Cancer |
| Date of Protocol: | |
| Version # 05 | October 08, 2014 |
| Version # 06 | November 20, 2014 |
| Version # 07 | January 26, 2015 |
| <b>Sponsor Contact:</b> | Altor BioScience |
| | Hing C. Wong, Ph.D. Altor Bioscience Corporation. Miramar, Florida 33025 Telephone: 954-443-8600 Safety Data Fax: 954-443-8602 |
| • • • | test that I have read, and that I understand and will abide by estrictions contained in the attached protocol. |
| Review Board (IRB), and I underst | is study without approval of the appropriate Institutional tand that any changes in the protocol must be approved in I, in certain cases the FDA, before they can be implemented, hazards to subjects. |
| Principal Investigator's Signature | Date |
| Principal Investigator's Name (Print) | ) |

Statistician: Study Coordinator: N/A

Zoe Moodie, PhD Fred Hutchinson Cancer Research Center 1100 Fairview Ave N, Mail Stop M2-C200 Seattle, WA 98109 (206) 667-7077 Fax: (206) 667-4378 zoe@fhcrc.org

Responsible Research Nurse: N/A Responsible Data Manager: N/A

NCI-Supplied Agent(s): N/A

Other Agent(s): ALT-803: a "recombinant human superagonist interleukin-15 (IL-15) complex" (AKA, IL-15N72D: IL-15RαSu/IgG1 Fc complex) NSC#: TBD

| <b>Investigational Agent</b> | IND# | IND Sponsor |
|------------------------------|--------|------------------------------|
| ALT-803 | 118280 | Altor Bioscience Corporation |

Protocol Type / Version # / Version Date: Amendment / Version 5.0 / January 21, 2015

### CANCER TRIALS SUPPORT UNIT (CTSU) ADDRESS AND CONTACT INFORMATION

| To submit site registration | For patient enrollments: | Submit study data |
|---|---|---|
| documents: | | |
| CTSU Regulatory Office<br>1818 Market Street, Suite 1100<br>Philadelphia, PA 19103<br>Phone – 1-866-651-CTSU | Please refer to the patient enrollment section for instructions on using the Oncology Patient Enrollment Network (OPEN) at | Data collection for this study will be done via Medidata Rave (Axio Research). |
| Fax – 215-569-0206 Email: CTSURegulatory@ctsu.coccg.o rg (for submitting regulatory documents only) | https://www.ctsu.org/OPEN_SYSTEM/ or https://OPEN.ctsu.org. Contact the CTSU Help Desk with any OPEN-related questions at ctsucontact@westat.com. | Please see the data submission section of the protocol for further instructions. |

The current version of the **study protocol and all supporting documents** must be downloaded from the protocol-specific Web page of the CTSU Member Web site located at <a href="https://www.ctsu.org">https://www.ctsu.org</a>.

## For patient eligibility or treatment-related questions:

Contact the CITN Coordinating Center at citn@fherc.org or 206-667-6606

For questions unrelated to patient eligibility, treatment, or clinical data submission contact the CTSU Help Desk by phone or e-mail:

CTSU General Information Line – 1-888-823-5923, or <a href="mailto:ctsucontact@westat.com">ctsucontact@westat.com</a>. All calls and correspondence will be triaged to the appropriate CTSU representative.

The CTSU Web site is located at <a href="https://www.ctsu.org">https://www.ctsu.org</a>

### **SCHEMA**

| | Regimen Description | | | | |
|---|---|---|---|---|---|
| Agent | Pre-Medications: Precautions | Dose | Route | Schedule | Cycle Length |
| ALT-803 | *1 dose of | $0.3 \mu\text{g/kg}$ or | IV | D1, W1 | 42 days |
| | antipyretic medication within | 0.5 μg/kg or<br>1 μg/kg or | | D1, W2 | (4 weeks on, 2 weeks off) |
| | 30 min of ALT-803 | $3 \mu g/kg$ or | | D1, W3 | With up to 4 cycles in the absence of unacceptable |
| | administration | 6 μg/kg | | D1, W4 | toxicity and disease |
| | *1 dose of | | | | progression** |
| | antipyretic | | | | |
| | medication 4 h after | | | | |
| | ALT-803 | | | | |
| | administration | | | | |

<sup>\*</sup>Non-steroidal anti-inflammatory medication including agents such as acetaminophen, ibuprofen, or Naproxen may be given per physician discretion. Not to exceed standard maximum thresholds:

Acetaminophen: not to exceed 3000 mg (3 g) in 24 hours

Ibuprofen: not to exceed 2400 mg in 24 hours Naproxen: not to exceed 1100 mg in 24 hours

<sup>\*\*</sup> Additional cycles beyond the 4<sup>th</sup> cycle may be considered for patients continuing to benefit and tolerating therapy, upon discussion among the sponsor and Principal Investigator.

| | Dose Escalation Schedule |
|------------|--------------------------------------------------|
| Dose Level | Dose of ALT-803 |
| Level -1 | 0.1 μg/kg (only if the first level is too toxic) |
| Level 1 | 0.3 μg/kg |
| Level 2 | 0.5 μg/kg |
| Level 3 | 1 μg/kg |
| Level 4 | 3 μg/kg |
| Level 5 | 6 μg/kg |

# 10. STUDY CALENDAR

Baseline evaluations are to be conducted within 1 to 30 days before start of protocol therapy, as indicated in the study calendar, except for pregnancy testing, which must be performed within 48 hours prior to initial ALT-803 administration. Scans and x-rays must be performed within 30 days before the start of therapy. In the event that the patient's condition is changing, laboratory evaluations should be repeated within 24 hours before initiating the next cycle of therapy. Please refer to the study calendar below for specific timing of required evaluations.

| | | 1. | | | | | | | | | | | | | | F/U | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Pre-s<br>(scree | | | | Cycle 1 | (Weeks) | | | | | Cycle | 2 (Weeks) | | | 14 d<br>post<br>last inf. | 6<br>Mo | 1 year <sup>i</sup> |
| | Within 30 d | Within<br>14 d | W1<br>D1±1 | W2<br>D8±1 | W3<br>D15±1 | W4<br>D22±1 | W5<br>D29±1 | W6<br>D36±1 | W1<br>D1±1 | W2<br>D8±1 | W3<br>D15±1 | W4<br>D22±1 | W5<br>D29±1 | W6<br>D36±1 | last IIII. | 1410 | 1 year |
| ALT-803*(A) | | | X | X | X | X | | | X | X | X | X | | | | | |
| Informed consent | X | | | | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | | | | | |
| Concomitant meds | X | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Physical exam <sup>h</sup> | | X | X | X | X | X | X | | X | X | X | X | X | | X | X | X |
| Vital signs with oxygen saturation | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Height | X | | | | | | | | | | | | | | | | |
| Weight | X | X | X | | X | | X | X | X | X | | X | | X | X | X | X |
| Performance status | | X | X | | | | | | X | | | | | | X | X | X |
| CBC w/diff, plts | | X | $X^k$ | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| PT/PTT | | X | | | | | | | | | | | | | | | |
| Serum chemistry <sup>a</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Antinuclear antibody (ANA) | X | | | | | | | | X | | | | | | | X | X |
| Electrocardiogram (ECG) <sup>b</sup> | | | X | X | X | X | | | X | X | X | X | | | X | X | X |
| ECHO (as indicated) | X | | | | | | | | | | | | | | | | |
| Adverse event evaluation | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Tumor measurements <sup>c</sup> CT, MRI, or PET of chest, abdomen, pelvis <sup>d</sup> | X<br>X | | Tumor measurements are repeated every $6 \pm 1$ week and $12 \pm 2$ weeks Documentation (radiologic) must be provided for patients removed from study for progressive disease. | | | | | | | | | | X | | | | |
| CT or MRI Brain <sup>d</sup> [as indicated for sympt only] | X | | | | | If negati | ve at base | eline, to b | e repeate | d only w | ith sympto | oms | | | | X | |

| | | | | | | | | | | | | | | | | F/U | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Pre-s<br>(scree | · | | | Cvela 1 | (Weeks) | | | | | Cycle | 2 (Weeks) | | | 14 d<br>post<br>last inf. | 6<br>Mo | 1 year <sup>i</sup> |
| | Within | Within | W1 | W2 | W3 | W4 | W5 | W6 | W1 | W2 | W3 | W4 | W5 | W6 | last IIII. | 1410 | 1 year |
| | 30 d | 14 d | D1±1 | D8±1 | D15±1 | D22±1 | D29±1 | D36±1 | D1±1 | | D15±1 | D22±1 | D29±1 | D36±1 | | | |
| Radiologic evaluation by RECIST 1.1 | Radiologic evaluation by X Radiologic measurements should be performed every $6 \pm 1$ week and $12 \pm 2$ weeks | | | | | | | | | | X | | | | | | |
| B-HCG <sup>e</sup> | | | X | | | | | | | | | | | | | | |
| Thyroid studies: TSH, T4 | X | | | | | | | | | | | | | | | X | X |
| PK <sup>f</sup> | | | X | | | | | | | | | | | | | | |
| WB Immunophenotyping <sup>g</sup> | | | X | X | X | X | X | | X | | X | | X | | | | |
| IFN-γ ELISPOT <sup>g</sup> | | | X | | | | X | | X | | | | X | | | | |
| NK-cell function <sup>g</sup> | | | X | | | | X | | X | | | | X | | | | |
| Plasma cytokines <sup>g</sup> | | | X | | | | X | | X | | | | X | | | | |
| Kyn/Trp ratio <sup>g</sup> | | | X | | | | X | | X | | | | X | | | | |
| Serum Ab to ALT-803 <sup>g</sup> | | | X | | | | | | X | | | | | | X | | |
| Other laboratories <sup>j</sup> | | | X | | | | | | | | | | | | | | |
| Serum | | | | | | | X | | X | | | | X | | | | |

Abbreviations: Ab, antibodies; CBC, complete blood count; CT, computed tomography; MRI, magnetic resonance imaging; NK, natural killer; PET, positron emission tomography; PK, pharmacokinetics; PTT, partial thromboplastin time; PT, prothrombin time

<sup>\*(</sup>A): Agent

<sup>&</sup>lt;sup>a</sup> Blood chemistries include: creatinine, glucose, total protein, blood urea nitrogen (BUN), total carbon dioxide (CO<sub>2</sub>), albumin, total bilirubin, phosphorus, alkaline phosphatase, aspartate transaminase (AST), and alanine transaminase (ALT)

<sup>&</sup>lt;sup>b</sup> ECGs are to be done before ALT-803 infusions on Day 1 and 4, 12 and 24 hours after the first ALT-803 infusion (Cycle 1, Week 1, Day1). As clinically indicated, ECGs are to be obtained to evaluate for cardiac toxicity during subsequent doses and cycles of therapy and follow-up visits.

<sup>&</sup>lt;sup>c</sup> Baseline tumor assessment scans should be done 1 to 30 days before beginning treatment.

<sup>&</sup>lt;sup>d</sup> CT, MRI, or PET is acceptable for imaging assessment purposes

<sup>&</sup>lt;sup>e</sup> Pregnancy test may be done up to 48 hours before ALT-803 administration

f See pharmacokinetic flow sheet for specific draw times

g Blood for WB Immunophenotyping, IFN-γ ELISPOT, NK-cell function, plasma cytokines, Kyn/Trp ratio and serum Ab to ALT-803 must be drawn **before** the patient receives ALT-803 infusions on Days 1, 8, 15, and 22 of each treatment cycle.

h Physical exam must always include neurological assessment. In addition, a funduscopic exam, conducted by the investigator with a hand-held ophthalmoscope, must be done prior to starting therapy (Cycle 1, Day 1, Week 1) and repeated if clinically indicated (See Section 6.0 for additional details).

<sup>&</sup>lt;sup>1</sup>Additional cycles beyond the 4<sup>th</sup> cycle may be considered for patients continuing to benefit and tolerating therapy, upon discussion among the sponsor and Principal Investigator. <sup>j</sup>Other labs include: Lactate dehydrogenase, magnesium, phosphate, CK and troponin I or T; must be drawn **before** and at 12 and 24 hours after the first ALT-803 dose. <sup>k</sup>CBC w/diff, plts (Cycle 1, Week 1, Day 1); must be drawn **before** and at **12** and **24** hours after the first ALT-803 dose.

Version Date: *June 11, 2015* 

NCI Protocol #: CITN-06-ALT-803

**Local Protocol #:** CA-ALT-803-01-13

**TITLE:** A Phase 1 Study of the Clinical and Immunologic Effects of ALT-803, a Novel Recombinant IL-15 Complex in Patients with Advanced Solid Tumors: Melanoma, Renal Cell, Non-Small Cell Lung and Squamous Cell Head and Neck Cancer

Sponsor: Alter BioScience

Hing C. Wong, Ph.D.

Altor Bioscience Corporation.

Miramar, Florida 33025

Telephone: 954-443-8600 Safety Data Fax: 954-443-8602

**Coordinating Center:** Cancer Immunotherapy Trials Network, Fred Hutchinson

Cancer Research Center

\*Principal Investigator: Marc Ernstoff, MD

Cleveland Clinic Foundation

9500 Euclid Avenue Cleveland, OH 44195

(216) 444-0888 ernstom@ccf.org

**Co-Investigators:** Lionel Lewis, MD

Dartmouth Hitchcock Medical Center

(603) 650-8685

lionel.lewis@dartmouth.edu

Sylvia Lee, MD

Seattle Cancer Care Alliance

(206) 667-2218 smlee@fhcrc.org

Shernan Holtan, MD University of Minnesota

(612) 301-1095 <u>sgholtan@umn.edu</u>

Version Date: *June 11, 2015* 

Howard L. Kaufman, MD, FACS Rutgers University (732) 235-6807 Howard.kaufman@rutgers.edu

Vamsidhar Velcheti, MD Cleveland Clinic Foundation (216) 444-8665 velchev@ccf.org

Thomas Waldmann, MD National Cancer Institute (301) 496-6656 tawald@mail.nih.gov

The SCCA, Cleveland Clinic Foundation, UCSF, University of Minnesota and Rutgers University will participate to the dose-escalation phase of the trial. NCI will be added in the expansion phase of the trial.

NCI Protocol #: CITN-06-ALT-803 Version Date: *June 11, 2015* 

# INVESTIGATOR SIGNATURE PAGE

| <b>Protocol Number:</b> | CA-ALT-803-01-13 |
|---|---|
| Protocol Title: | A Phase 1 Study of the Clinical and<br>Immunologic Effects of ALT-803, a Novel<br>Recombinant IL-15 Complex in Patients with<br>Advanced Solid Tumors: Melanoma, Renal Cell,<br>Non-Small Cell Lung and Squamous Cell Head<br>and Neck Cancer |
| Date of Protocol: | |
| Version # 05 | October 08, 2014 |
| Version # 06 | November 20, 2014 |
| Version # 07 | January 26, 2015 |
| Version #08 | June 11, 2015 |
| <b>Sponsor Contact:</b> | Altor BioScience |
| | Hing C. Wong, Ph.D. |
| | Altor Bioscience Corporation. |
| | Miramar, Florida 33025 |
| | Telephone: 954-443-8600 |
| | Safety Data Fax: 954-443-8602 |
| all the conditions, instructions, and re<br>Additionally, I will not initiate thi<br>Review Board (IRB), and I underst | est that I have read, and that I understand and will abide by estrictions contained in the attached protocol. s study without approval of the appropriate Institutional and that any changes in the protocol must be approved in , in certain cases the FDA, before they can be implemented, hazards to subjects. |
| Principal Investigator's Signature | Date |
| Principal Investigator's Name (Print) | |

Version Date: *June 11, 2015* 

Statistician: Study Coordinator: N/A

Zoe Moodie, PhD Fred Hutchinson Cancer Research Center 1100 Fairview Ave N, Mail Stop M2-C200 Seattle, WA 98109 (206) 667-7077 Fax: (206) 667-4378

zoe@fhcrc.org

Responsible Research Nurse: N/A Responsible Data Manager: N/A

NCI-Supplied Agent(s): N/A

Other Agent(s): ALT-803: a "recombinant human superagonist interleukin-15 (IL-15) complex"

(AKA, IL-15N72D: IL-15RαSu/IgG1 Fc complex) NSC#: TBD

| Investigational Agent | IND# | IND Sponsor |
|-----------------------|--------|------------------------------|
| ALT-803 | 118280 | Altor Bioscience Corporation |

Protocol Type / Version # / Version Date: Amendment / Version 6.0 / June 3, 2015

Version Date: *June 11, 2015* 

# CANCER TRIALS SUPPORT UNIT (CTSU) ADDRESS AND CONTACT INFORMATION

| To submit site registration | For patient enrollments: | Submit study data |
|---|---|---|
| documents: | | |
| CTSU Regulatory Office | Please refer to the patient enrollment | Data collection for this |
| 1818 Market Street, Suite 1100 | section for instructions on using the | study will be done via |
| Philadelphia, PA 19103 | Oncology Patient Enrollment Network | Medidata Rave (Axio |
| Phone – 1-866-651-CTSU | (OPEN) at | Research). |
| Fax – 215-569-0206 | https://www.ctsu.org/OPEN_SYSTEM/ | |
| Email: | or <a href="https://OPEN.ctsu.org">https://OPEN.ctsu.org</a> . | Please see the data |
| CTSURegulatory@ctsu.coccg.o | | submission section of the |
| rg (for submitting regulatory | Contact the CTSU Help Desk with any | protocol for further |
| documents only) | OPEN-related questions at | instructions. |
| | ctsucontact@westat.com. | |

The current version of the **study protocol and all supporting documents** must be downloaded from the protocol-specific Web page of the CTSU Member Web site located at <a href="https://www.ctsu.org">https://www.ctsu.org</a>.

# For patient eligibility or treatment-related questions:

Contact the CITN Coordinating Center at citn@fhcrc.org or 206-667-6606

For questions unrelated to patient eligibility, treatment, or clinical data submission contact the CTSU Help Desk by phone or e-mail:

CTSU General Information Line – 1-888-823-5923, or <u>ctsucontact@westat.com</u>. All calls and correspondence will be triaged to the appropriate CTSU representative.

The CTSU Web site is located at <a href="https://www.ctsu.org">https://www.ctsu.org</a>

Version Date: *June 11, 2015* 

### **SCHEMA**

| | Regimen Description | | | | |
|---|---|---|---|---|---|
| Agent | Pre-Medications: Precautions | Dose | Route | Schedule | Cycle Length |
| ALT-803 | *1 dose of | 0.3 μg/kg or | IV | D1, W1 | 42 days |
| | antipyretic medication within | 0.5 μg/kg or<br>1 μg/kg or | | D1, W2 | (4 weeks on, 2 weeks off) With up to 4 cycles in the |
| | 30 min of ALT-803<br>administration | 3 μg/kg or<br>6 μg/kg | | D1, W3<br>D1, W4 | absence of unacceptable toxicity and disease |
| | *1 dose of<br>antipyretic<br>medication 4 h after<br>ALT-803<br>administration | | | | progression** |

<sup>\*</sup>Non-steroidal anti-inflammatory medication including agents such as acetaminophen, ibuprofen, or Naproxen may be given per physician discretion. Not to exceed standard maximum thresholds:

Acetaminophen: not to exceed 3000 mg (3 g) in 24 hours

Ibuprofen: not to exceed 2400 mg in 24 hours Naproxen: not to exceed 1100 mg in 24 hours

<sup>\*\*</sup> Additional cycles beyond the 4<sup>th</sup> cycle may be considered for patients continuing to benefit and tolerating therapy, upon discussion among the sponsor and Principal Investigator.

| | Dose Escalation Schedule |
|---|---|
| Dose Level | Dose of ALT-803 |
| Level -1 | 0.1 μg/kg (only if the first level is too toxic) |
| Level 1 | 0.3 μg/kg |
| Level 2 | 0.5 μg/kg |
| Level 3 | 1 μg/kg |
| Level 4 | 3 μg/kg |
| Level 5 | 6 μg/kg |

Version Date: *June 11, 2015* 

## 10. STUDY CALENDAR

Baseline evaluations are to be conducted within 1 to 30 days before start of protocol therapy, as indicated in the study calendar, except for pregnancy testing, which must be performed within 48 hours prior to initial ALT-803 administration. Scans and x-rays must be performed within 30 days before the start of therapy. In the event that the patient's condition is changing, laboratory evaluations should be repeated within 24 hours before initiating the next cycle of therapy. Please refer to the study calendar below for specific timing of required evaluations.

| | | | | | | | | | | | | | | | | | | T/U | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | study<br>ening) | | | Сус | cle 1 (We | eeks) | | | | Cycle 2 (Weeks) | | | | 14 days<br>post last<br>infusion | 6<br>Mo | 1<br>year <sup>i</sup> | | |
| | Within<br>30 days | Within<br>14 days | We<br>D1±1 | ek 1<br><b>D4±1</b> | W2<br>D8±1 | W3<br>D15±1 | W4<br>D22±1 | W5<br>D29±1 | W6<br>D36±1 | We<br>D1±1 | ek 1<br><b>D4</b> ±1 | W2<br>D8±1 | W3<br>D15±1 | W4<br>D22±1 | W5<br>D29±1 | W6<br>D36±1 | | | |
| ALT-803*(A) | 30 days | 14 days | X | D4±1 | X | X | X | D29±1 | D30±1 | X | D4±1 | X | X | X | D29±1 | D30±1 | | | - |
| Informed consent | X | | | | | | | | | | | | | | | | | | <u> </u> |
| Demographics | X | | | | | | | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | | | | | | | |
| Concomitant meds | X | | X | | X | X | X | X | X | X | | X | X | X | X | X | X | X | X |
| Physical exam <sup>h</sup> | | X | X | | X | X | X | X | | X | | X | X | X | X | | X | X | X |
| Vital signs with oxygen saturation | | X | X | | X | X | X | X | X | X | | X | X | X | X | X | X | X | X |
| Height | X | | | | | | | | | | | | | | | | | | |
| Weight | X | X | X | | | X | | X | X | X | | X | | X | | X | X | X | X |
| Performance status | | X | X | | | | | | | X | | | | | | | X | X | X |
| CBC w/diff, plts | | X | $X^k$ | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| PT/PTT | | X | | | | | | | | | | | | | | | | | |
| Serum chemistry <sup>a</sup> | | X | X | | X | X | X | X | X | X | | X | X | X | X | X | X | X | X |
| Antinuclear antibody (ANA) | X | | | | | | | | | X | | | | | | | | X | X |
| Electrocardiogram (ECG) <sup>b</sup> | | | X | | X | X | X | | | X | | X | X | X | | | X | X | X |
| ECHO (as indicated) | X | | | | | | | | | | | | | | | | | | |
| Adverse event evaluation | | X | X | | X | X | X | X | X | X | | X | X | X | X | X | X | X | X |
| Tumor measurements <sup>c</sup> | X | | | <b>I</b> | | Tumor n | neasuren | ents are | repeated | every 6 = | ± 1 week | and 12 = | ± 2 weeks | S . | | l | <u> </u> | X | 1 |
| CT, MRI, or PET of chest, abdomen, pelvis <sup>d</sup> | X | | Tumor measurements are repeated every $6 \pm 1$ week and $12 \pm 2$ weeks Documentation (radiologic) must be provided for patients removed from study for progressive disease. | | | | | | | | | | | | | | | | |
| CT or MRI Brain <sup>d</sup> [as indicated for sympt only] | X | | If negative at baseline, to be repeated only with symptoms | | | | | | | | | | X | | | | | | |
| Radiologic evaluation by RECIST 1.1 | X | | | | Radio | logic me | asuremen | nts should | d be perfo | ormed ev | ery 6 ± 1 | week a | nd 12 ± 2 | weeks | | | | X | |

Version Date: *June 11, 2015* 

| | | | | | | | | | | | | | | | | | F | T/U | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | study<br>ening) | | | Сус | ele 1 (We | eks) | | | | Cycle 2 (Weeks) | | | | 14 days<br>post last<br>infusion | 6<br>Mo | 1<br>year <sup>i</sup> | | |
| | Within 30 days | Within<br>14 days | We<br>D1±1 | ek 1<br><b>D4</b> ±1 | W2<br>D8±1 | W3<br>D15±1 | W4<br>D22±1 | W5<br>D29±1 | W6<br>D36±1 | We<br>D1±1 | ek 1<br><b>D4±1</b> | W2<br>D8±1 | W3<br>D15±1 | W4<br>D22±1 | W5<br>D29±1 | W6<br>D36±1 | | | |
| B-HCG <sup>e</sup> | 20 44.75 | 1. 44.75 | X | 2 | 20-1 | B10=1 | D22-1 | 527-1 | 250-1 | | 2,-1 | 20-1 | B10-1 | D22-1 | 527-1 | 200-1 | | | |
| Thyroid studies: TSH, T4 | X | | | | | | | | | | | | | | | | | X | X |
| PK <sup>f</sup> | | | X | | | | | | | | | | | | | | | | |
| WB Immunophenotyping <sup>g</sup> | | | X | X | X | X | X | X | | X | X | | | | X | | | | |
| IFN-γ ELISPOT <sup>g</sup> | | | X | | | | | X | | X | | | | | | | | | |
| NK-cell function <sup>g</sup> | | | X | X | X | | | X | | X | X | | | | | | | | |
| Plasma cytokines <sup>g</sup> | | | X | | | | | X | | X | | | | | X | | | | |
| Kyn/Trp ratio <sup>g</sup> | | | X | | | | | X | | X | | | | | X | | | | |
| Serum Ab to ALT-803 <sup>g</sup> | | | X | | | | | | | X | | | | | | | X | | |
| Other laboratories <sup>j</sup> | | | X | | | | | | | | | | | | | | | | |
| Serum Storage (optional) | | | X | | | | | X | | | | | | | | | | | |

Abbreviations: Ab, antibodies; CBC, complete blood count; CT, computed tomography; MRI, magnetic resonance imaging; NK, natural killer; PET, positron emission tomography; PK, pharmacokinetics; PTT, partial thromboplastin time; PT, prothrombin time

<sup>\*(</sup>A): Agent

<sup>&</sup>lt;sup>a</sup> Blood chemistries include: creatinine, glucose, total protein, blood urea nitrogen (BUN), total carbon dioxide (CO<sub>2</sub>), albumin, total bilirubin, phosphorus, alkaline phosphatase, aspartate transaminase (AST), and alanine transaminase (ALT)

<sup>&</sup>lt;sup>b</sup> ECGs are to be done before ALT-803 infusions on Day 1 and 4, 12 and 24 hours after the first ALT-803 infusion (Cycle 1, Week 1, Day1). As clinically indicated, ECGs are to be obtained to evaluate for cardiac toxicity during subsequent doses and cycles of therapy and follow-up visits.

<sup>&</sup>lt;sup>c</sup> Baseline tumor assessment scans should be done 1 to 30 days before beginning treatment.

<sup>&</sup>lt;sup>d</sup> CT, MRI, or PET is acceptable for imaging assessment purposes

e Pregnancy test may be done up to 48 hours before ALT-803 administration

f See pharmacokinetic flow sheet for specific draw times

g Blood for WB Immunophenotyping, IFN-γ ELISPOT, NK-cell function, plasma cytokines, Kyn/Trp ratio and serum Ab to ALT-803 must be drawn **before** the patient receives ALT-803 infusions on Days 1, 8, 15, and 22 of each treatment cycle.

h Physical exam must always include neurological assessment. In addition, a funduscopic exam, conducted by the investigator with a hand-held ophthalmoscope, must be done prior to starting therapy (Cycle 1, Day 1, Week 1) and repeated if clinically indicated (See Section 6.0 for additional details).

Additional cycles beyond the 4th cycle may be considered for patients continuing to benefit and tolerating therapy, upon discussion among the sponsor and Principal Investigator.

<sup>&</sup>lt;sup>j</sup>Other labs include: Lactate dehydrogenase, magnesium, phosphate, CK and troponin I or T; must be drawn **before** and at 12 and 24 hours after the first ALT-803 dose.

<sup>&</sup>lt;sup>k</sup>CBC w/diff, plts (Cycle 1, Week 1, Day 1); must be drawn **before** and at **12** and **24** hours after the first ALT-803 dose.

NCI Protocol #: CITN-06-ALT-803

**Local Protocol #:** CA-ALT-803-01-13

**TITLE:** A Phase 1 Study of the Clinical and Immunologic Effects of ALT-803, a Novel Recombinant IL-15 Complex in Patients with Advanced Solid Tumors: Melanoma, Renal Cell, Non-Small Cell Lung and Squamous Cell Head and Neck Cancer

Sponsor: Alter BioScience

Hing C. Wong, Ph.D.

Altor Bioscience Corporation.

Miramar, Florida 33025

Telephone: 954-443-8600 Safety Data Fax: 954-443-8602

**Coordinating Center:** Cancer Immunotherapy Trials Network, Fred Hutchinson

Cancer Research Center

\*Principal Investigator: Marc Ernstoff, MD

Cleveland Clinic Foundation

9500 Euclid Avenue Cleveland, OH 44195

(216) 444-0888 ernstom@ccf.org

Co-Investigators: Lionel Lewis, MD

Dartmouth Hitchcock Medical Center

(603) 650-8685

lionel.lewis@dartmouth.edu

Sylvia Lee, MD

Seattle Cancer Care Alliance

(206) 667-2218 smlee@fhcrc.org

Shernan Holtan, MD University of Minnesota

(612) 301-1095 <u>sgholtan@umn.edu</u>

> Howard L. Kaufman, MD, FACS Rutgers University (732) 235-6807 Howard.kaufman@rutgers.edu

Vamsidhar Velcheti, MD Cleveland Clinic Foundation (216) 444-8665 velchev@ccf.org

Thomas Waldmann, MD National Cancer Institute (301) 496-6656 tawald@mail.nih.gov

The SCCA, Cleveland Clinic Foundation, UCSF, University of Minnesota and Rutgers University will participate to the dose-escalation phase of the trial. NCI will be added in the expansion phase of the trial.

# INVESTIGATOR SIGNATURE PAGE

| <b>Protocol Number:</b> | CA-ALT-803-01-13 |
|---|---|
| Protocol Title: | A Phase 1 Study of the Clinical and<br>Immunologic Effects of ALT-803, a Novel<br>Recombinant IL-15 Complex in Patients with<br>Advanced Solid Tumors: Melanoma, Renal Cell,<br>Non-Small Cell Lung and Squamous Cell Head<br>and Neck Cancer |
| Date of Protocol: | |
| Version # 05 | October 08, 2014 |
| Version # 06 | November 20, 2014 |
| Version # 07 | January 26, 2015 |
| Version # 08 | June 11, 2015 |
| Version # 09 | August 5, 2015 |
| <b>Sponsor Contact:</b> | Altor BioScience |
| | Hing C. Wong, Ph.D. |
| | Altor Bioscience Corporation. |
| | Miramar, Florida 33025 |
| | Telephone: 954-443-8600 |
| | Safety Data Fax: 954-443-8602 |
| | test that I have read, and that I understand and will abide by restrictions contained in the attached protocol. |
| Review Board (IRB), and I underst | is study without approval of the appropriate Institutional tand that any changes in the protocol must be approved in I, in certain cases the FDA, before they can be implemented, hazards to subjects. |
| Principal Investigator's Signature | Date |
| Principal Investigator's Name (Print | <u>)</u> |

Statistician: Study Coordinator: N/A

Zoe Moodie, PhD Fred Hutchinson Cancer Research Center 1100 Fairview Ave N, Mail Stop M2-C200 Seattle, WA 98109 (206) 667-7077 Fax: (206) 667-4378

zoe@fhcrc.org

Responsible Research Nurse: N/A Responsible Data Manager: N/A

NCI-Supplied Agent(s): N/A

Other Agent(s): ALT-803: a "recombinant human superagonist interleukin-15 (IL-15) complex" (AKA, IL-15N72D: IL-15RαSu/IgG1 Fc complex) NSC#: TBD

| Investigational Agent | IND# | IND Sponsor |
|-----------------------|--------|------------------------------|
| ALT-803 | 118280 | Altor Bioscience Corporation |

Protocol Type / Version # / Version Date: Amendment / Version 7.0 / July 28, 2015

## CANCER TRIALS SUPPORT UNIT (CTSU) ADDRESS AND CONTACT INFORMATION

| To submit site registration | For patient enrollments: | Submit study data |
|---|---|---|
| documents: | | |
| CTSU Regulatory Office<br>1818 Market Street, Suite 1100<br>Philadelphia, PA 19103<br>Phone – 1-866-651-CTSU | Please refer to the patient enrollment section for instructions on using the Oncology Patient Enrollment Network (OPEN) at | Data collection for this study will be done via Medidata Rave (Axio Research). |
| Fax – 215-569-0206 Email: CTSURegulatory@ctsu.coccg.o rg (for submitting regulatory documents only) | https://www.ctsu.org/OPEN_SYSTEM/ or https://OPEN.ctsu.org. Contact the CTSU Help Desk with any OPEN-related questions at ctsucontact@westat.com. | Please see the data submission section of the protocol for further instructions. |

The current version of the **study protocol and all supporting documents** must be downloaded from the protocol-specific Web page of the CTSU Member Web site located at <a href="https://www.ctsu.org">https://www.ctsu.org</a>.

# For patient eligibility or treatment-related questions:

Contact the CITN Coordinating Center at citn@fherc.org or 206-667-6606

For questions unrelated to patient eligibility, treatment, or clinical data submission contact the CTSU Help Desk by phone or e-mail:

CTSU General Information Line – 1-888-823-5923, or <a href="mailto:ctsucontact@westat.com">ctsucontact@westat.com</a>. All calls and correspondence will be triaged to the appropriate CTSU representative.

The CTSU Web site is located at <a href="https://www.ctsu.org">https://www.ctsu.org</a>

#### **SCHEMA**

| | Regimen Description | | | | |
|---|---|---|---|---|---|
| Agent | Pre-Medications: Precautions | Dose | Route | Schedule | Cycle Length |
| ALT-803 | *1 dose of | 0.3 μg/kg or | IV | D1, W1 | 42 days |
| | antipyretic medication within | 0.5 μg/kg or<br>1 μg/kg or | | D1, W2 | (4 weeks on, 2 weeks off) |
| | 30 min of ALT-803 | 3 μg/kg or | | D1, W3 | With up to 4 cycles in the absence of unacceptable |
| | administration | 6 μg/kg | | D1, W4 | toxicity and disease |
| | *1 dose of<br>antipyretic<br>medication 4 h after<br>ALT-803<br>administration | 6 μg/kg<br>10 μg/kg<br>15 μg/kg<br>20 μg/kg | SQ | | progression** |

<sup>\*</sup>Non-steroidal anti-inflammatory medication including agents such as acetaminophen, ibuprofen, or Naproxen may be given per physician discretion. Not to exceed standard maximum thresholds:

Acetaminophen: not to exceed 3000 mg (3 g) in 24 hours

Ibuprofen: not to exceed 2400 mg in 24 hours Naproxen: not to exceed 1100 mg in 24 hours

<sup>\*\*</sup> Additional cycles beyond the 4<sup>th</sup> cycle may be considered for patients continuing to benefit and tolerating therapy, upon discussion among the sponsor and Principal Investigator.

| Dose Escalation Schedule | | |
|---|---|---|
| Dose Level | Dose of ALT-803 | Route of Administration |
| Level -1 | 0.1 μg/kg (only if the first level is too toxic) | |
| Level 1 | 0.3 μg/kg | IV |
| Level 2 | 0.5 μg/kg | <i>IV</i> |
| Level 3 | 1 μg/kg | <i>IV</i> |
| Level 4 | 3 μg/kg | <i>IV</i> |
| Level 5 | 6 μg/kg | <i>IV</i> |
| Level 5a <sup>1</sup> | 6 μg/kg | SQ |
| Level 6 | 10 μg/kg | SQ |
| Level 7 | 15 μg/kg | SQ |
| Level 8 <sup>2</sup> | 20 μg/kg | SQ |

<sup>&</sup>lt;sup>1</sup>With protocol version #9, ALT-803 dosing is changed from IV to SQ, and dose level 5 is repeated to confirm safety with the new route of administration.

<sup>&</sup>lt;sup>2</sup>The dose of ALT-803 will be increased in increments of 5 μg/kg if a minimum of three patients have been treated at dose level 8 (20 μg/kg), and the Maximum Tolerated Dose (MTD) and Optimum Biological Dose (OBD) have not been identified. Enrollment will continue until the MTD/OBD is identified.

## 10. STUDY CALENDAR

Baseline evaluations are to be conducted within 1 to 30 days before start of protocol therapy, as indicated in the study calendar, except for pregnancy testing, which must be performed within 48 hours prior to initial ALT-803 administration. Scans and x-rays must be performed within 30 days before the start of therapy. In the event that the patient's condition is changing, laboratory evaluations should be repeated within 24 hours before initiating the next cycle of therapy. Please refer to the study calendar below for specific timing of required evaluations.

| | | | | | | | | | | | | | | | | | | T/U | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | study<br>ening) | | | Cvc | ele 1 (We | eks) | | | | | Cvo | cle 2 (We | eks) | | | 14 days<br>post last<br>dose | 6<br>Mo | 1<br>vear <sup>i</sup> |
| | Within | Within | We | | W2 | W3 | W4 | W5 | W6 | We | | W2 | W3 | W4 | W5 | W6 | | | <i>J</i> • |
| ALT-803*(A) | 30 days | 14 days | D1±1<br>X | D4±1 | D8±1<br>X | D15±1 | D22±1<br>X | D29±1 | D36±1 | D1±1<br>X | D4±1 | D8±1<br>X | D15±1 | D22±1<br>X | D29±1 | D36±1 | | $\vdash$ | |
| Informed consent | X | | | | | | | | | | | | | | | | | $\vdash$ | |
| Demographics | X | | | | | | | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | | | | | | | |
| Concomitant meds | X | | X | | X | X | X | X | X | X | | X | X | X | X | X | X | X | X |
| Physical exam <sup>h</sup> | | X | X | | X | X | X | X | | X | | X | X | X | X | | X | X | X |
| Vital signs with oxygen saturation | | X | X | | X | X | X | X | X | X | | X | X | X | X | X | X | X | X |
| Height | X | | | | | | | | | | | | | | | | | | |
| Weight | X | X | X | | | X | | X | X | X | | X | | X | | X | X | X | X |
| Performance status | | X | X | | | | | | | X | | | | | | | X | X | X |
| CBC w/diff, plts | | X | X <sup>k</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| PT/PTT | | X | | | | | | | | | | | | | | | | | |
| Serum chemistry <sup>a</sup> | | X | X | | X | X | X | X | X | X | | X | X | X | X | X | X | X | X |
| Antinuclear antibody (ANA) | X | | | | | | | | | X | | | | | | | | X | X |
| Electrocardiogram (ECG) <sup>b</sup> | | | X | | X | X | X | | | X | | X | X | X | | | X | X | X |
| ECHO (as indicated) | X | | | | | | | | | | | | | | | | | | |
| Adverse event evaluation | | X | X | | X | X | X | X | X | X | | X | X | X | X | X | X | X | X |
| Tumor measurements <sup>c</sup> | X | | Tumor measurements are repeated every $6 \pm 1$ week and $12 \pm 2$ weeks | | | | | | | | | | X | | | | | | |
| CT, MRI, or PET of chest, abdomen, pelvis <sup>d</sup> | X | | Documentation (radiologic) must be provided for patients removed from study for progressive disease. | | | | | | | | | | | | | | | | |
| CT or MRI Brain <sup>d</sup> [as indicated for sympt only] | X | | If negative at baseline, to be repeated only with symptoms | | | | | | | | | | X | | | | | | |
| Radiologic evaluation by RECIST 1.1 | X | | Radiologic measurements should be performed every $6 \pm 1$ week and $12 \pm 2$ weeks | | | | | | | | | X | | | | | | | |

| | Poss | -4 J | | | | | | | | | | | | | | | 14 days | /U | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | study<br>ening) | | | Cvc | ele 1 (We | eks) | | | | | Cyc | ele 2 (We | eks) | | | post last<br>dose | 6<br>Mo | l<br>vear <sup>i</sup> |
| | Within | Within | We | ek 1 | W2 | W3 | W4 | W5 | W6 | We | ek 1 | W2 | W3 | W4 | W5 | W6 | uose | 1110 | year |
| | 30 days | 14 days | D1±1 | D4±1 | D8±1 | D15±1 | D22±1 | D29±1 | D36±1 | D1±1 | D4±1 | D8±1 | D15±1 | D22±1 | D29±1 | D36±1 | | | |
| Injection Site Evaluation | | | | X | X | X | X | | | X | X | X | X | X | | | X | | |
| B-HCG <sup>e</sup> | | | X | | | | | | | | | | | | | | | | |
| Thyroid studies: TSH, T4 | X | | | | | | | | | | | | | | | | | X | X |
| PK <sup>f</sup> | | | X | | | | | | | | | | | | | | | | |
| WB Immunophenotyping <sup>g</sup> | | | X | X | X | X | X | X | | X | X | | | | X | | | | |
| IFN-γ ELISPOT <sup>g</sup> | | | X | | | | | X | | X | | | | | | | | | |
| NK-cell function <sup>g</sup> | | | X | X | X | | | X | | X | X | | | | | | | | |
| Plasma cytokines <sup>g</sup> | | | X | | | | | X | | X | | | | | X | | | | |
| Kyn/Trp ratio <sup>g</sup> | | | X | | | | | X | | X | | | | | X | | | | |
| Serum Ab to ALT-803 <sup>g</sup> | | | X | | | | | | | X | | | | | | | X | | |
| Other laboratories <sup>j</sup> | | | X | | | | | | | | | | | | | | | | |
| Serum Storage (optional) | | | X | | | | | X | | | | | | | | | | | |

Abbreviations: Ab, antibodies; CBC, complete blood count; CT, computed tomography; MRI, magnetic resonance imaging; NK, natural killer; PET, positron emission tomography; PK, pharmacokinetics; PTT, partial thromboplastin time; PT, prothrombin time

<sup>\*(</sup>A): Agent

<sup>&</sup>lt;sup>a</sup> Blood chemistries include: creatinine, glucose, total protein, blood urea nitrogen (BUN), total carbon dioxide (CO<sub>2</sub>), albumin, total bilirubin, phosphorus, alkaline phosphatase, aspartate transaminase (AST), and alanine transaminase (ALT)

<sup>&</sup>lt;sup>b</sup> ECGs are to be done before ALT-803 *administration* on Day 1 and 4, 12 and 24 hours after the first ALT-803 *dose* (Cycle 1, Week 1, Day1). As clinically indicated, ECGs are to be obtained to evaluate for cardiac toxicity during subsequent doses and cycles of therapy and follow-up visits.

<sup>&</sup>lt;sup>c</sup> Baseline tumor assessment scans should be done 1 to 30 days before beginning treatment.

<sup>&</sup>lt;sup>d</sup> CT, MRI, or PET is acceptable for imaging assessment purposes

<sup>&</sup>lt;sup>e</sup> Pregnancy test may be done up to 48 hours before ALT-803 administration

f See pharmacokinetic flow sheet for specific draw times

g Blood for WB Immunophenotyping, IFN-γ ELISPOT, NK-cell function, plasma cytokines, Kyn/Trp ratio and serum Ab to ALT-803 must be drawn **before** the patient receives *the dose of* ALT-803 on Days 1, 8, 15, and 22 of each treatment cycle.

h Physical exam must always include neurological assessment. In addition, a funduscopic exam, conducted by the investigator with a hand-held ophthalmoscope, must be done prior to starting therapy (Cycle 1, Day 1, Week 1) and repeated if clinically indicated (See Section 6.0 for additional details).

Additional cycles beyond the 4<sup>th</sup> cycle may be considered for patients continuing to benefit and tolerating therapy, upon discussion among the sponsor and Principal Investigator.

<sup>&</sup>lt;sup>j</sup>Other labs include: Lactate dehydrogenase, magnesium, phosphate, CK and troponin I or T; must be drawn **before** and at 12 and 24 hours after the first ALT-803 dose.

<sup>&</sup>lt;sup>k</sup>CBC w/diff, plts (Cycle 1, Week 1, Day 1); must be drawn **before** and at **12** and **24** hours after the first ALT-803 dose.

Version Date: April 13, 2016

NCI Protocol #: CITN-06-ALT-803

**Local Protocol #:** CA-ALT-803-01-13

**TITLE:** A Phase 1 Study of the Clinical and Immunologic Effects of ALT-803, a Novel Recombinant IL-15 Complex in Patients with Advanced Solid Tumors: Melanoma, Renal Cell, Non-Small Cell Lung and Squamous Cell Head and Neck Cancer

Sponsor: Alter BioScience

Hing C. Wong, Ph.D.

Altor Bioscience Corporation.

Miramar, Florida 33025

Telephone: 954-443-8600 Safety Data Fax: 954-443-8602

**Coordinating Center:** Cancer Immunotherapy Trials Network, Fred Hutchinson

Cancer Research Center

\*Principal Investigator: Marc Ernstoff, MD

Roswell Park Cancer Institute

Elm & Carlton Streets Buffalo, NY 14263 (716) 845-4101

marc.ernstoff@roswellpark.org

Co-Principal Investigator: Kim Margolin, MD

City of Hope (626) 218-0496 kmargolin@coh.org

Co-Investigators: Lionel Lewis, MD

Dartmouth Hitchcock Medical Center

(603) 650-8685

lionel.lewis@dartmouth.edu

Sylvia Lee, MD

Seattle Cancer Care Alliance

(206) 667-2218 smlee@fhcrc.org

Shernan Holtan, MD


University of Minnesota (612) 301-1095 sgholtan@umn.edu

Howard L. Kaufman, MD, FACS Rutgers University (732) 235-6807 Howard.kaufman@rutgers.edu

Vamsidhar Velcheti, MD Cleveland Clinic Foundation (216) 444-8665 velchev@ccf.org

Thomas Waldmann, MD National Cancer Institute (301) 496-6656 tawald@mail.nih.gov

The SCCA, Cleveland Clinic Foundation, UCSF, University of Minnesota and Rutgers University will participate to the dose-escalation phase of the trial. NCI will be added in the expansion phase of the trial.


# INVESTIGATOR SIGNATURE PAGE

| <b>Protocol Number:</b> | CA-ALT-803-01-13 |
|---|---|
| Protocol Title: | A Phase 1 Study of the Clinical and<br>Immunologic Effects of ALT-803, a Novel<br>Recombinant IL-15 Complex in Patients with<br>Advanced Solid Tumors: Melanoma, Renal Cell,<br>Non-Small Cell Lung and Squamous Cell Head<br>and Neck Cancer |
| Date of Protocol: | |
| Version # 05 | October 08, 2014 |
| Version # 06 | November 20, 2014 |
| Version # 07 | January 26, 2015 |
| Version # 08 | June 11, 2015 |
| Version # 09 | August 5, 2015 |
| Version # 10 | April 13, 2016 |
| <b>Sponsor Contact:</b> | Altor BioScience |
| | Hing C. Wong, Ph.D. |
| | Altor Bioscience Corporation. |
| | Miramar, Florida 33025 |
| | Telephone: 954-443-8600 |
| | Safety Data Fax: 954-443-8602 |
| , , , | est that I have read, and that I understand and will abide by estrictions contained in the attached protocol. |
| Review Board (IRB), and I underst | is study without approval of the appropriate Institutional and that any changes in the protocol must be approved in , in certain cases the FDA, before they can be implemented, hazards to subjects. |
| Principal Investigator's Signature | Date |
| 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 | |
| Principal Investigator's Name (Print) | |


Statistician:

Study Coordinator: N/A

Zoe Moodie, PhD Fred Hutchinson Cancer Research Center 1100 Fairview Ave N, Mail Stop M2-C200 Seattle, WA 98109

(206) 667-7077

Fax: (206) 667-4378

zoe@fhcrc.org

Responsible Research Nurse: N/A Responsible Data Manager: N/A

NCI-Supplied Agent(s): N/A

Other Agent(s): ALT-803: a "recombinant human superagonist interleukin-15 (IL-15) complex"

(AKA, IL-15N72D: IL-15RαSu/IgG1 Fc complex) NSC#: TBD

| <b>Investigational Agent</b> | IND# | IND Sponsor |
|------------------------------|--------|------------------------------|
| ALT-803 | 118280 | Altor Bioscience Corporation |

Protocol Type / Version # / Version Date: Amendment / Version 8.0 / March 31, 2016


### CANCER TRIALS SUPPORT UNIT (CTSU) ADDRESS AND CONTACT INFORMATION

| To submit site registration | For patient enrollments: | Submit study data |
|---|---|---|
| documents: | | |
| CTSU Regulatory Office | Please refer to the patient enrollment | Data collection for this |
| 1818 Market Street, Suite 1100 | section for instructions on using the | study will be done via |
| Philadelphia, PA 19103 | Oncology Patient Enrollment Network | Medidata Rave (Axio |
| Phone – 1-866-651-CTSU | (OPEN) at | Research). |
| Fax – 215-569-0206 | https://www.ctsu.org/OPEN_SYSTEM/ | · |
| Email: | or <a href="https://OPEN.ctsu.org">https://OPEN.ctsu.org</a> . | Please see the data |
| CTSURegulatory@ctsu.coccg.o | | submission section of the |
| rg (for submitting regulatory | Contact the CTSU Help Desk with any | protocol for further |
| documents only) | OPEN-related questions at | instructions. |
| • , | ctsucontact@westat.com. | |

The current version of the **study protocol and all supporting documents** must be downloaded from the protocol-specific Web page of the CTSU Member Web site located at <a href="https://www.ctsu.org">https://www.ctsu.org</a>.

# For patient eligibility or treatment-related questions:

Contact the CITN Coordinating Center at citn@fhcrc.org or 206-667-6606

For questions unrelated to patient eligibility, treatment, or clinical data submission contact the CTSU Help Desk by phone or e-mail:

CTSU General Information Line – 1-888-823-5923, or <a href="mailto:ctsucontact@westat.com">ctsucontact@westat.com</a>. All calls and correspondence will be triaged to the appropriate CTSU representative.

The CTSU Web site is located at <a href="https://www.ctsu.org">https://www.ctsu.org</a>


### **SCHEMA**

| Regimen Description | | | | | |
|---|---|---|---|---|---|
| Agent | Pre-Medications: Precautions | Dose | Route | Schedule | Cycle Length |
| ALT-803 | *1 dose of | 0.3 μg/kg or | IV | D1, W1 | 42 days |
| | antipyretic<br>medication within<br>30 min of ALT-803<br>administration | 0.5 μg/kg or<br>1 μg/kg or<br>3 μg/kg or<br>6 μg/kg | | D1, W2<br>D1, W3 | (4 weeks on, 2 weeks of With up to 4 cycles in the absence of unacceptable |
| | *1 dose of<br>antipyretic<br>medication 4 h after<br>ALT-803<br>administration | 6 μg/kg<br>10 μg/kg<br>15 μg/kg<br>20 μg/kg | SQ | D1, W4 | toxicity and disease progression** |

<sup>\*</sup>Non-steroidal anti-inflammatory medication including agents such as acetaminophen, ibuprofen, or Naproxen may be given per physician discretion. Not to exceed standard maximum thresholds:

Acetaminophen: not to exceed 3000 mg (3 g) in 24 hours

Ibuprofen: not to exceed 2400 mg in 24 hours Naproxen: not to exceed 1100 mg in 24 hours

<sup>\*\*</sup> Additional cycles beyond the 4<sup>th</sup> cycle may be considered for patients continuing to benefit and tolerating therapy, upon discussion among the sponsor and Principal Investigator.

| Dose Escalation Schedule | | |
|---|---|---|
| Dose Level | Dose of ALT-803 | Route of Administration |
| Level -1 | 0.1 μg/kg (only if the first level is too toxic) | IV |
| Level 1 | 0.3 μg/kg | IV |
| Level 2 | 0.5 μg/kg | IV |
| Level 3 | 1 μg/kg | IV |
| Level 4 | 3 μg/kg | IV |
| Level 5 | 6 μg/kg | IV |
| Level 5a <sup>1</sup> | 6 μg/kg | SQ |
| Level 6 | 10 μg/kg | SQ |
| Level 7 | 15 μg/kg | SQ |
| Level 8 <sup>2</sup> | 20 μg/kg | SQ |

<sup>&</sup>lt;sup>1</sup>With protocol version #9, ALT-803 dosing is changed from IV to SQ, and dose level 5 is repeated to confirm safety with the new route of administration.

 $<sup>^2</sup>$ The dose of ALT-803 will be increased in increments of 5 µg/kg if a minimum of three patients have been treated at dose level 8 (20 µg/kg), and the Maximum Tolerated Dose (MTD) and Optimum Biological Dose (OBD) have not been identified. Enrollment will continue until the MTD/OBD is identified.


## 10. STUDY CALENDAR

Baseline evaluations are to be conducted within 1 to 30 days before start of protocol therapy, as indicated in the study calendar, except for pregnancy testing, which must be performed within 48 hours prior to initial ALT-803 administration. Scans and x-rays must be performed within 30 days before the start of therapy. In the event that the patient's condition is changing, laboratory evaluations should be repeated within 24 hours before initiating the next cycle of therapy. Please refer to the study calendar below for specific timing of required evaluations.

| | | | | | | | | | | | | | | | | | F | F/U | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | study<br>ening) | | | Cyc | ele 1 (We | eks) | | | | | Cyc | cle 2 (We | eeks) | | | 14 days<br>post last<br>dose | 6<br>Mo | 1<br>year <sup>i</sup> |
| | Within<br>30 days | Within<br>14 days | We<br>D1±1 | ek 1<br><b>D4</b> ±1 | W2<br>D8±1 | W3<br>D15±1 | W4<br>D22±1 | W5<br>D29±1 | W6<br>D36±1 | We<br>D1±1 | ek 1<br><b>D4</b> ±1 | W2<br>D8±1 | W3<br>D15±1 | W4<br>D22±1 | W5<br>D29±1 | W6<br>D36±1 | | | |
| ALT-803*(A) | 30 days | 14 days | X | D4±1 | X | X | X | D29±1 | D30±1 | X | D4±1 | X | X | X | D29±1 | D30±1 | | | - |
| Informed consent | X | | | | | | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | | | | | | | |
| Concomitant meds | X | | X | | X | X | X | X | X | X | | X | X | X | X | X | X | X | X |
| Physical exam <sup>h</sup> | | X | X | | X | X | X | X | | X | | X | X | X | X | | X | X | X |
| Vital signs with oxygen saturation | | X | X | | X | X | X | X | X | X | | X | X | X | X | X | X | X | X |
| Height | X | | | | | | | | | | | | | | | | | | |
| Weight | X | X | X | | | X | | X | X | X | | X | | X | | X | X | X | X |
| Performance status | | X | X | | | | | | | X | | | | | | | X | X | X |
| CBC w/diff, plts | | X | $X^k$ | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| PT/PTT | | X | | | | | | | | | | | | | | | | | |
| Serum chemistry <sup>a</sup> | | X | X | | X | X | X | X | X | X | | X | X | X | X | X | X | X | X |
| Antinuclear antibody (ANA) | X | | | | | | | | | X | | | | | | | | X | X |
| Electrocardiogram (ECG) <sup>b</sup> | | | X | | X | X | X | | | X | | X | X | X | | | X | X | X |
| ECHO (as indicated) | X | | | | | | | | | | | | | | | | | | |
| Adverse event evaluation | | X | X | | X | X | X | X | X | X | | X | X | X | X | X | X | X | X |
| Tumor measurements <sup>c</sup> | X | | Tumor measurements are repeated every $6 \pm 1$ week and $12 \pm 2$ weeks | | | | | | | | | I | X | | | | | | |
| CT, MRI, or PET of chest, abdomen, pelvis <sup>d</sup> | X | | Documentation (radiologic) must be provided for patients removed from study for progressive disease. | | | | | | | | | | | | | | | | |
| CT or MRI Brain <sup>d</sup> [as indicated for sympt only] | X | | If negative at baseline, to be repeated only with symptoms | | | | | | | | | X | | | | | | | |
| Radiologic evaluation by RECIST 1.1 | X | | Radiologic measurements should be performed every $6 \pm 1$ week and $12 \pm 2$ weeks | | | | | | | | | X | | | | | | | |


| | | | | | | | | | | | | | | | | | | F/U | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Pre- | study | | | | | | | | | | | | | | | 14 days<br>post last | 6 | 1 |
| | (scre | ening) | | | Cyc | ele 1 (We | eks) | | | | | Cyc | le 2 (We | eks) | | | dose | Mo | yeari |
| | Within | Within | Wee | ek 1 | W2 | W3 | W4 | W5 | W6 | We | ek 1 | W2 | W3 | W4 | W5 | W6 | | | |
| | 30 days | 14 days | D1±1 | D4±1 | D8±1 | D15±1 | D22±1 | D29±1 | D36±1 | D1±1 | D4±1 | D8±1 | D15±1 | D22±1 | D29±1 | D36±1 | | | |
| Injection Site Evaluation | | | | X | X | X | X | | | X | X | X | X | X | | | X | | |
| B-HCG <sup>e</sup> | | | X | | | | | | | | | | | | | | | | |
| Thyroid studies: TSH, T4 | X | | | | | | | | | | | | | | | | | X | X |
| PK <sup>f</sup> | | | X | | | | | | | | | | | | | | | | |
| WB Immunophenotyping <sup>g</sup> | | | X | X | X | X | X | X | | X | X | | | | X | | | | |
| IFN-γ ELISPOT <sup>g</sup> | | | X | | | | | X | | X | | | | | | | | | |
| NK-cell function <sup>g</sup> | | | X | X | X | | | X | | X | X | | | | | | | | |
| Plasma cytokines <sup>g</sup> | | | X | | | | | X | | X | | | | | X | | | | |
| Kyn/Trp ratio <sup>g</sup> | | | X | | | | | X | | X | | | | | X | | | | |
| Serum Ab to ALT-803 <sup>g</sup> | | | X | | | | | | | X | | | | | | | X | | |
| Other laboratories <sup>j</sup> | | | X | | | | | | | | | | | | | | | | |
| Serum Storage (optional) | | | X | | | | | X | | | | | | | | | | | |

Abbreviations: Ab, antibodies; CBC, complete blood count; CT, computed tomography; MRI, magnetic resonance imaging; NK, natural killer; PET, positron emission tomography; PK, pharmacokinetics; PTT, partial thromboplastin time; PT, prothrombin time

<sup>\*(</sup>A): Agent

<sup>&</sup>lt;sup>a</sup> Blood chemistries include: creatinine, glucose, total protein, blood urea nitrogen (BUN), total carbon dioxide (CO<sub>2</sub>), albumin, total bilirubin, phosphorus, alkaline phosphatase, aspartate transaminase (AST), and alanine transaminase (ALT)

<sup>&</sup>lt;sup>b</sup> ECGs are to be done before ALT-803 *administration* on Day 1 and 4, 12 and 24 hours after the first ALT-803 *dose* (Cycle 1, Week 1, Day1). As clinically indicated, ECGs are to be obtained to evaluate for cardiac toxicity during subsequent doses and cycles of therapy and follow-up visits.

<sup>&</sup>lt;sup>c</sup> Baseline tumor assessment scans should be done 1 to 30 days before beginning treatment.

<sup>&</sup>lt;sup>d</sup> CT, MRI, or PET is acceptable for imaging assessment purposes

<sup>&</sup>lt;sup>e</sup> Pregnancy test may be done up to 48 hours before ALT-803 administration

f See pharmacokinetic flow sheet for specific draw times

g Blood for WB Immunophenotyping, IFN-γ ELISPOT, NK-cell function, plasma cytokines, Kyn/Trp ratio and serum Ab to ALT-803 must be drawn **before** the patient receives *the dose of* ALT-803 on Days 1, 8, 15, and 22 of each treatment cycle.

h Physical exam must always include neurological assessment. In addition, a funduscopic exam, conducted by the investigator with a hand-held ophthalmoscope, must be done prior to starting therapy (Cycle 1, Day 1, Week 1) and repeated if clinically indicated (See Section 6.0 for additional details).

Additional cycles beyond the 4<sup>th</sup> cycle may be considered for patients continuing to benefit and tolerating therapy, upon discussion among the sponsor and Principal Investigator.

<sup>&</sup>lt;sup>j</sup>Other labs include: Lactate dehydrogenase, magnesium, phosphate, CK and troponin I or T; must be drawn **before** and at 12 and 24 hours after the first ALT-803 dose.

<sup>&</sup>lt;sup>k</sup>CBC w/diff, plts (Cycle 1, Week 1, Day 1); must be drawn **before** and at **12** and **24** hours after the first ALT-803 dose.

NCI Protocol #: CITN-06-ALT-803

**Local Protocol #:** CA-ALT-803-01-13

**TITLE:** A Phase 1 Study of the Clinical and Immunologic Effects of ALT-803, a Novel Recombinant IL-15 Complex in Patients with Advanced Solid Tumors: Melanoma, Renal Cell, *Sarcoma, Colon, Non-Hodgkin Lymphoma*, Non-Small Cell Lung and Squamous Cell Head and Neck Cancer *and Cutaneous Squamous Cell Cancer* 

Sponsor: Alter BioScience

Hing C. Wong, Ph.D.

Altor Bioscience Corporation.

Miramar, Florida 33025

Telephone: 954-443-8600 Safety Data Fax: 954-443-8602

**Coordinating Center:** Cancer Immunotherapy Trials Network, Fred Hutchinson

Cancer Research Center

\*Principal Investigator: Marc Ernstoff, MD

Roswell Park Cancer Institute

Elm & Carlton Streets Buffalo, NY 14263 (716) 845-4101

marc.ernstoff@roswellpark.org

Co-Principal Investigator: Kim Margolin, MD

City of Hope (626) 218-0496 kmargolin@coh.org

Jeffrey S. Miller

University of Minnesota

(612) 625-7409 <u>Mille011@umn.edu</u>

Co-Investigators: Lionel Lewis, MD

Dartmouth Hitchcock Medical Center

(603) 650-8685

lionel.lewis@dartmouth.edu

> Sylvia Lee, MD Seattle Cancer Care Alliance (206) 667-2218 smlee@fhcrc.org

Shernan Holtan, MD University of Minnesota (612) 301-1095 sgholtan@umn.edu

Howard L. Kaufman, MD, FACS Rutgers University (732) 235-6807 Howard.kaufman@rutgers.edu

Vamsidhar Velcheti, MD Cleveland Clinic Foundation (216) 444-8665 velchev@ccf.org

Thomas Waldmann, MD National Cancer Institute (301) 496-6656 tawald@mail.nih.gov

The SCCA, Cleveland Clinic Foundation, University of Minnesota and Rutgers University will participate to the dose-escalation phase of the trial. NCI will be added in the expansion phase of the trial.

# INVESTIGATOR SIGNATURE PAGE

| <b>Protocol Number:</b> | CA-ALT-803-01-13 |
|---|---|
| Protocol Title: | A Phase 1 Study of the Clinical and Immunologic Effects of ALT-803, a Novel Recombinant IL-15 Complex in Patients with Advanced Solid Tumors: Melanoma, Renal Cell, <i>Sarcoma, Colon, Non-Hodgkin Lymphoma,</i> Non-Small Cell Lung and Squamous Cell Head and Neck Cancer and <i>Cutaneous Squamous Cell Cancer</i> |
| Date of Protocol: | |
| Version # 05 | October 08, 2014 |
| Version # 06 | November 20, 2014 |
| Version # 07 | January 26, 2015 |
| Version # 08 | June 11, 2015 |
| Version # 09 | August 5, 2015 |
| Version # 11 | August 9, 2016 |
| <b>Sponsor Contact:</b> | Altor BioScience |
| | Hing C. Wong, Ph.D. |
| | Altor Bioscience Corporation. |
| | Miramar, Florida 33025 |
| | Telephone: 954-443-8600 |
| | Safety Data Fax: 954-443-8602 |
| | attest that I have read, and that I understand and will abide by and restrictions contained in the attached protocol. |
| Review Board (IRB), and I und | this study without approval of the appropriate Institutional terstand that any changes in the protocol must be approved in and, in certain cases the FDA, before they can be implemented, ate hazards to subjects. |
| Principal Investigator's Signature | Date |
| Principal Investigator's Name (Pr | rint) |

Statistician: Study Coordinator: N/A

Zoe Moodie, PhD Fred Hutchinson Cancer Research Center 1100 Fairview Ave N, Mail Stop M2-C200 Seattle, WA 98109 (206) 667-7077

Fax: (206) 667-4378 zoe@fhcrc.org

Responsible Research Nurse: N/A Responsible Data Manager: N/A

NCI-Supplied Agent(s): N/A

Other Agent(s): ALT-803: a "recombinant human superagonist interleukin-15 (IL-15) complex" (AKA, IL-15N72D: IL-15RαSu/IgG1 Fc complex) NSC#: TBD

| <b>Investigational Agent</b> | IND# | IND Sponsor |
|------------------------------|--------|------------------------------|
| ALT-803 | 118280 | Altor Bioscience Corporation |

Protocol Type / Version # / Version Date: Amendment 9 / Version 2.0 / July 13, 2016

### CANCER TRIALS SUPPORT UNIT (CTSU) ADDRESS AND CONTACT INFORMATION

| To submit site registration documents: | For patient enrollments: | Submit study data |
|---|---|---|
| CTSU Regulatory Office 1818 Market Street, Suite 1100 Philadelphia, PA 19103 Phone – 1-866-651-CTSU Fax – 215-569-0206 Email: CTSURegulatory@ctsu.coccg.o rg (for submitting regulatory documents only) | Please refer to the patient enrollment section for instructions on using the Oncology Patient Enrollment Network (OPEN) at <a href="https://www.ctsu.org/OPEN_SYSTEM/">https://www.ctsu.org/OPEN_SYSTEM/</a> or <a href="https://OPEN.ctsu.org">https://OPEN.ctsu.org</a> . Contact the CTSU Help Desk with any OPEN-related questions at ctsucontact@westat.com. | Data collection for this study will be done via Medidata Rave (Axio Research). Please see the data submission section of the protocol for further instructions. |

The current version of the **study protocol and all supporting documents** must be downloaded from the protocol-specific Web page of the CTSU Member Web site located at <a href="https://www.ctsu.org">https://www.ctsu.org</a>.

# For patient eligibility or treatment-related questions:

Contact the CITN Coordinating Center at <a href="mailto:citn@fhcrc.org">citn@fhcrc.org</a> or 206-667-6606

For questions unrelated to patient eligibility, treatment, or clinical data submission contact the CTSU Help Desk by phone or e-mail:

CTSU General Information Line – 1-888-823-5923, or <a href="mailto:ctsucontact@westat.com">ctsucontact@westat.com</a>. All calls and correspondence will be triaged to the appropriate CTSU representative.

The CTSU Web site is located at <a href="https://www.ctsu.org">https://www.ctsu.org</a>

### **SCHEMA**

| | | Regimen D | Description | 1 | |
|---|---|---|---|---|---|
| Agent | Pre-Medications: Precautions | Dose | Route | Schedule | Cycle Length |
| ALT-803 | *1 dose of<br>antipyretic<br>medication within<br>30 min of ALT-803<br>administration | 0.3 μg/kg or<br>0.5 μg/kg or<br>1 μg/kg or<br>3 μg/kg or<br>6 μg/kg | IV<br>SQ | D1, W1<br>D1, W2<br>D1, W3<br>D1, W4 | 42 days (4 weeks on, 2 weeks off) With up to 4 cycles in the absence of unacceptable toxicity and disease progression** |
| | *1 dose of antipyretic medication 4 h after ALT-803 administration | 10 μg/kg<br>15 μg/kg<br>20 μg/kg | 54 | | Progression |
| | | 10 μg/kg +<br>15 μg/kg SQ<br>15 μg/kg +<br>15 μg/kg SQ<br>20 μg/kg +<br>15 μg/kg SQ | IT<br>followed<br>by SQ | D1, W1<br>(IT)<br>D1, W2<br>(SQ)<br>D1, W3<br>(SQ)<br>D1, W4<br>(SQ) | 42 days (4 weeks on, 2 weeks off) With up to 4 cycles in the absence of unacceptable toxicity and disease progression** Cycle 1 only: pre and post treatment biopsy |

<sup>\*</sup>Non-steroidal anti-inflammatory medication including agents such as acetaminophen, ibuprofen, or Naproxen may be given per physician discretion. Not to exceed standard maximum thresholds:

Acetaminophen: not to exceed 3000 mg (3 g) in 24 hours

Ibuprofen: not to exceed 2400 mg in 24 hours Naproxen: not to exceed 1100 mg in 24 hours

\*\* Additional cycles beyond the 4<sup>th</sup> cycle may be considered for patients continuing to benefit and tolerating therapy, upon discussion among the sponsor and Principal Investigator.

| | Dose Escalation Schedule | |
|---|---|---|
| | Cohort 1 | |
| Dose Level | Dose of ALT-803 | Route of Administration |
| Level -1 | 0.1 μg/kg (only if the first level is too toxic) | IV |
| Level 1 | 0.3 μg/kg | IV |
| Level 2 | 0.5 μg/kg | IV |
| Level 3 | 1 μg/kg | IV |
| Level 4 | 3 μg/kg | IV |
| Level 5 | 6 μg/kg | IV |
| | Cohort 2 <sup>3</sup> | |

| Level 5a <sup>1</sup> | 6 μg/kg | SQ |
|-----------------------|-------------------------|-------------------|
| Level 6 | 10 μg/kg | SQ |
| Level 7 | 15 μg/kg | SQ |
| Level 8 <sup>2</sup> | 20 μg/kg | SQ |
| · | Cohort 3 <sup>3,4</sup> | |
| Level 1 | 10 μg/kg | IT (Week 1) |
| Level 1 | 15 μg/kg | SQ (Week 2, 3, 4) |
| Level 2 | 15 μg/kg | IT (Week 1) |
| Level 2 | 15 μg/kg | SQ (Week 2, 3, 4) |
| Level 3 <sup>2</sup> | 20 μg/kg | IT (Week 1) |
| Level 3 | 15 μg/kg | SQ (Week 2, 3, 4) |

<sup>&</sup>lt;sup>1</sup>With protocol version #9, ALT-803 dosing is changed from IV to SQ, and dose level 5 is repeated to confirm safety with the new route of administration.

<sup>&</sup>lt;sup>2</sup>The dose of ALT-803 will be increased in increments of 5 μg/kg if a minimum of three patients have been treated at dose level 8 *in Cohort 2 or dose level 3 in Cohort 3*, and the Maximum Tolerated Dose (MTD) and Optimum Biological Dose (OBD) have not been identified. Enrollment will continue until the MTD/OBD is identified.

<sup>&</sup>lt;sup>3</sup>Cohort 2 and Cohort 3 enrollment will occur in parallel. The treatment cohort assignment (Cohort 2 vs Cohort 3) is at the Investigator and patient discretion. Cohort 3 will be receiving both IT injection and SQ injections and must be amenable to undergoing pre and post-treatment biopsy.

<sup>&</sup>lt;sup>4</sup>Cohort 3, dose escalation only for the IT portion; SQ dose remains constant at 15 μg/kg.

## 10. STUDY CALENDAR

Baseline evaluations are to be conducted within 1 to 30 days before start of protocol therapy, as indicated in the study calendar, except for pregnancy testing, which must be performed within 48 hours prior to initial ALT-803 administration. Scans and x-rays must be performed within 30 days before the start of therapy. In the event that the patient's condition is changing, laboratory evaluations should be repeated within 24 hours before initiating the next cycle of therapy. Please refer to the study calendar below for specific timing of required evaluations.

| | | | | | | | | | | | | | | | | | | T/U | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | study<br>ening) | | | Cvo | ele 1 (We | eks) | | | | | 14 days<br>post last<br>dose | 6<br>Mo | 1<br>vear <sup>i</sup> | | | | | |
| | Within | Within | We | | W2 | W3 | W4 | W5 | W6 | We | | W2 | W3 | W4 | W5 | W6 | | | 3 |
| ALT-803 | 30 days | 14 days | D1±1<br>X <sup>l</sup> | D4±1 | D8±1<br>X | D15±1 | D22±1<br>X | D29±1 | D36±1 | D1±1<br>X <sup>l</sup> | D4±1 | D8±1 | D15±1 | D22±1<br>X | D29±1 | D36±1 | | <del> </del> | |
| Informed consent | X | | 71 | | Λ | <i>A</i> | <i>A</i> | | | Α. | | A | 74 | 74 | | | | | |
| Demographics | X | | | | | | | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | | | | | | | |
| Concomitant meds | X | | X | | X | X | X | X | X | X | | X | X | X | X | X | X | X | X |
| Physical exam <sup>h</sup> | | X | X | | X | X | X | X | | X | | X | X | X | X | | X | X | X |
| Vital signs with oxygen saturation | | X | X | | X | X | X | X | X | X | | X | X | X | X | X | X | X | X |
| Height | X | | | | | | | | | | | | | | | | | | |
| Weight | X | X | X | | | X | | X | X | X | | X | | X | | X | X | X | X |
| Performance status | | X | X | | | | | | | X | | | | | | | X | X | X |
| CBC w/diff, plts | | X | $X^k$ | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| PT/PTT | | X | | | | | | | | | | | | | | | | | |
| Serum chemistry <sup>a</sup> | | X | X | | X | X | X | X | X | X | | X | X | X | X | X | X | X | X |
| Antinuclear antibody (ANA) | X | | | | | | | | | X | | | | | | | | X | X |
| Electrocardiogram (ECG) <sup>b</sup> | | | X | | X | X | X | | | X | | X | X | X | | | X | X | X |
| ECHO (as indicated) | X | | | | | | | | | | | | | | | | | | |
| Adverse event evaluation | | X | X | | X | X | X | X | X | X | | X | X | X | X | X | X | X | X |
| Tumor measurements <sup>c</sup> | X | | I | | I | Tumor n | neasurem | ents are | repeated | every 6 = | ± 1 week | and 12 = | ± 2 weeks | S | | | I | X | |
| CT, MRI, or PET of chest, abdomen, pelvis <sup>d</sup> | X | | | Docum | entation | (radiolog | gic) must | be provi | ded for p | atients re | emoved f | rom stuc | ly for pro | gressive | disease. | | | | |
| CT or MRI Brain <sup>d</sup> [as indicated for sympt only] | X | | | | | | | | ne, to be | • | | | | | | | | X | |
| Radiologic evaluation by RECIST 1.1 | X | | | | Radio | logic mea | asuremer | its should | l be perfo | ormed ev | $ery 6 \pm 1$ | week a | nd 12 ± 2 | weeks | | | | X | |

| | | | | | | | | | | | | | | | | | F | F/U | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | study<br>ening) | | | | | | | | | Cycle 2 (Weeks) | | | | | | | | 1<br>year <sup>i</sup> |
| | Within | Within | We | | W2 | W3 | W4 | W5 | W6 | | ek 1 | W2 | W3 | W4 | W5 | W6 | | Mo | |
| Injection Site Evaluation | 30 days | 14 days | D1±1 | <i>D4±1</i> X | D8±1<br>X | D15±1 | D22±1<br>X | D29±1 | D36±1 | D1±1<br>X | <i>D4±1</i> X | D8±1<br>X | D15±1 | D22±1<br>X | D29±1 | D36±1 | X | | |
| B-HCG <sup>e</sup> | | | X | | | | | | | | | | | | | | | | |
| Thyroid studies: TSH, T4 | X | | | | | | | | | | | | | | | | | X | X |
| PK <sup>f</sup> | | | X | | | | | | | | | | | | | | | | |
| WB Immunophenotyping <sup>g</sup> | | | X | X | X | X | X | X | | X | X | | | | X | | | | |
| IFN-γ ELISPOT <sup>g</sup> | | | X | | | | | X | | X | | | | | | | | | |
| NK-cell function <sup>g</sup> | | | X | X | X | | | X | | X | X | | | | | | | | |
| Plasma cytokines <sup>g</sup> | | | X | | | | | X | | X | | | | | X | | | | |
| Kyn/Trp ratio <sup>g</sup> | | | X | | | | | X | | X | | | | | X | | | | |
| Serum Ab to ALT-803g | | | X | | | | | | | X | | | | | | | X | | |
| Other laboratories <sup>j</sup> | | | X | | | | | | | | | | | | | | | | |
| Serum Storage (optional) | | | X | X | | | | | | | | | | | | | | | |
| Biopsy <sup>m</sup> | 1 | | X | | X | | | | | | | | | | | | | | |

Abbreviations: Ab, antibodies; CBC, complete blood count; CT, computed tomography; MRI, magnetic resonance imaging; NK, natural killer; PET, positron emission tomography; PK, pharmacokinetics; PTT, partial thromboplastin time; PT, prothrombin time

<sup>&</sup>lt;sup>a</sup> Blood chemistries include: creatinine, glucose, total protein, blood urea nitrogen (BUN), total carbon dioxide (CO<sub>2</sub>), albumin, total bilirubin, phosphorus, alkaline phosphatase, aspartate transaminase (AST), and alanine transaminase (ALT)

<sup>&</sup>lt;sup>b</sup> ECGs are to be done before ALT-803 *administration* on Day 1 and 4, 12 and 24 hours after the first ALT-803 *dose* (Cycle 1, Week 1, Day1). As clinically indicated, ECGs are to be obtained to evaluate for cardiac toxicity during subsequent doses and cycles of therapy and follow-up visits.

<sup>&</sup>lt;sup>c</sup> Baseline tumor assessment scans should be done 1 to 30 days before beginning treatment.

<sup>&</sup>lt;sup>d</sup> CT, MRI, or PET is acceptable for imaging assessment purposes

e Pregnancy test may be done up to 48 hours before ALT-803 administration

f See pharmacokinetic flow sheet for specific draw times

<sup>&</sup>lt;sup>g</sup> Blood for WB Immunophenotyping, IFN-γ ELISPOT, NK-cell function, plasma cytokines, Kyn/Trp ratio and serum Ab to ALT-803 must be drawn **before** the patient receives *the dose of* ALT-803 on Days 1, 8, 15, and 22 of each treatment cycle.

h Physical exam must always include neurological assessment. In addition, a funduscopic exam, conducted by the investigator with a hand-held ophthalmoscope, must be done prior to starting therapy (Cycle 1, Day 1, Week 1) and repeated if clinically indicated (See Section 6.0 for additional details).

Additional cycles beyond the 4th cycle may be considered for patients continuing to benefit and tolerating therapy, upon discussion among the sponsor and Principal Investigator.

Other labs include: Lactate dehydrogenase, magnesium, phosphate, CK and troponin I or T; must be drawn before and at 12 and 24 hours after the first ALT-803 dose.

<sup>\*</sup>CBC w/diff, plts (Cycle 1, Week 1, Day 1); must be drawn **before** and at **12** and **24** hours after the first ALT-803 dose.

<sup>&</sup>lt;sup>1</sup>Cohort 3 only, intratumoral injection (Week 1, Day 1 of each treatment cycle)

<sup>&</sup>lt;sup>m</sup>Cohort 3 only, biopsy must be done before ALT-803 administration